CLINICAL TRIAL: NCT03596762
Title: A Double-Blind, Randomised, Placebo Controlled, Adaptive Design Study of the Efficacy, Safety and Pharmacokinetics of NT-814 in Female Subjects With Moderate to Severe Vasomotor Symptoms Associated With the Menopause
Brief Title: A Study of BAY3427080 (NT-814) in the Treatment of Moderate to Severe Post-menopausal Vasomotor Symptoms
Acronym: SWITCH-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Nerre Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21686; 2018-002763-26 (EudraCT Number)
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Menopause; Hot Flashes; Night Waking
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 160 mg Elinzanetant (BAY3427080) (Experimental): Participants received 4x40 mg elinzanetant capsules.
  Interventions: Drug: Elinzanetant (BAY3427080)
- 120 mg Elinzanetant (BAY3427080) (Experimental): Participants received 3x40 mg elinzanetant capsules and 1 placebo capsule.
  Interventions: Drug: Elinzanetant (BAY3427080)
- 80 mg Elinzanetant (BAY3427080) (Experimental): Participants received 2x40 mg elinzanetant capsules and 2 placebo capsules.
  Interventions: Drug: Elinzanetant (BAY3427080)
- 40 mg Elinzanetant (BAY3427080) (Experimental): Participants received one 40 mg elinzanetant capsule and 3 placebo capsules.
  Interventions: Drug: Elinzanetant (BAY3427080)
- Placebo (Placebo Comparator): Participants received four placebo capsules orally once daily in the evening before bedtime.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — BAY3427080 capsules
  Other Names: NT-814
  Arms: 120 mg Elinzanetant (BAY3427080); 160 mg Elinzanetant (BAY3427080); 40 mg Elinzanetant (BAY3427080); 80 mg Elinzanetant (BAY3427080)
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of BAY3427080 (NT-814), taken once a day, in the treatment of troublesome post-menopausal symptoms.

DETAILED DESCRIPTION:
This is a multi-centre, multi-country, double-blind, randomised, placebo-controlled Phase 2b study. The study will have a single-blind run-in period and will be adaptive with respect to the number of subjects recruited into each dose group. Four doses of BAY3427080 (40 mg once a day, 80 mg once a day, 120 mg once a day and 160 mg once a day) will be investigated and compared to placebo, in five parallel groups. Subjects will participate in the study for a total of approximately 19 weeks, comprising a screening period of 1 week, a 14 week treatment period, and then a final follow up visit 4 weeks after the end of the treatment period. There will be a total of 8 visits whilst participating in the study. Subjects will record their hot flashes in an electronic diary during the screening period to establish eligibility and throughout the study after randomisation.

ELIGIBILITY:
Key Inclusion Criteria:

* Postmenopausal
* Body mass index between 18 and 38 kg/m2, inclusive
* Subject experiences moderate or severe hot flashes

Key Exclusion Criteria:

* Inability to comply with the use of prohibited and allowed medications as described in the protocol.
* Any prior or ongoing history of clinically relevant drug or alcohol abuse within 12 months of Screening.
* Any clinically significant prior or ongoing history of arrhythmias, either determined through clinical history or on ECG evaluation.
* Any clinically significant abnormal laboratory test result(s) measured at Screening.
* Any active ongoing condition that could have caused difficulty in interpreting vasomotor symptoms.
* Uncontrolled hypertension.
* A history or hyperthyroidism, hypothyroidism or abnormal thyroid function tests at Screening. Treated hypothyroidism with normal thyroid function test results at Screening is acceptable.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (10):
  - Study Site 12, Mesa, Arizona
  - Study Site 19, San Diego, California
  - Study Site 13, Aventura, Florida
  - Study Site 15, Lake Worth, Florida
  - Study Site 18, Atlanta, Georgia
  - Study Site 16, New Orleans, Louisiana
  - Study Site 10, Boston, Massachusetts
  - Study Site 11, Boston, Massachusetts
  - Study Site 17, Las Vegas, Nevada
  - Study Site 14, Houston, Texas
- Canada (5):
  - Study Site 50, Red Deer, Alberta
  - Study Site 51, Mission, British Columbia
  - Study Site 54, Guelph, Ontario
  - Study Site 52, Scarborough Village, Ontario
  - Study Site 53, Toronto, Ontario
- United Kingdom (10):
  - Study Site 37, Blackpool
  - Study Site 34, Cannock
  - Study Site 31, Glasgow
  - Study Site 39, Leeds
  - Study Site 38, Liverpool
  - Study Site 30, London
  - Study Site 36, Manchester
  - Study Site 33, Poole
  - Study Site 32, Southport
  - Study Site 35, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 20 November 2018 (first participant, first visit) and 21 November 2019 (last participant, last visit) at 11 sites in the USA, nine sites in the UK, and five sites in Canada.
Pre-assignment Details: A total of 760 participants were screened, of whom 199 completed screening and were randomised. Not meeting the eligibility criteria was the reason provided for all screening failures (561). A total of 47 participants were randomised to placebo and 152 participants to elinzanetant (BAY3427080).
Period: Overall Study
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Started | 47 | 31 | 17 | 52 | 52
Completed | 43 | 30 | 16 | 51 | 45
Not Completed | 4 | 1 | 1 | 1 | 7
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 5
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080) | Total
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (4.1) | 55.4 (4.0) | 55.9 (4.2) | 54.8 (4.4) | 55.0 (3.8) | 55.1 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 31 | 17 | 52 | 52 | 199
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 2 | 6 | 13
  Not Hispanic or Latino | 45 | 29 | 16 | 50 | 46 | 186
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 3 | 13 | 11 | 38
  White | 38 | 24 | 13 | 37 | 40 | 152
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Mean Daily Frequency of Moderate and Severe Hot Flushes From Baseline to Week 4
Description: Participants recorded daily in their electronic diary (eDiary) the frequency and severity of hot flushes during the treatment period. The baseline assessment for hot flushes was calculated using the last 7 days (not necessarily consecutive days) with an available data in the evening and/or the morning of the baseline diary completion period. A diary day was comprised of the evening entry of this day and the morning entry of the following day, in that order. Mean daily frequency = Sum of number of hot flushes filled in the diary during the last 7 diary days (with at least one available data in the evening and/or morning) divided by 7. Moderate: Sensation of heat with sweating, but able to continue activity. Severe: Sensation of heat with sweating, causing cessation (stopping) of activity.
Time Frame: From baseline to Week 4
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot flushes per day
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Hot flushes per day
  Baseline | 11.82 (4.42) | 12.13 (8.81) | 14.55 (5.87) | 13.54 (7.17) | 12.92 (6.90)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 52 | 47
  Week 4: Change from baseline | -2.45 (3.65) | -4.19 (5.78) | -4.30 (6.45) | -6.76 (5.85) | -5.42 (5.36)
Statistical Analysis 1: Comparison: Placebo vs 40 mg Elinzanetant (BAY3427080); Change from Baseline to Week 4; Test type: Superiority; p = 0.1946, Mixed-Effect Model Repeated Measures; Difference in LS means = -1.52, 95% CI 2-sided [-3.83 to 0.78]
Statistical Analysis 2: Comparison: Placebo vs 80 mg Elinzanetant (BAY3427080); Change from Baseline to Week 4; Test type: Superiority; p = 0.3682, Mixed-Effect Model Repeated Measures; Difference in LS means = 1.29, 95% CI 2-sided [-4.11 to 1.53]
Statistical Analysis 3: Comparison: Placebo vs 120 mg Elinzanetant (BAY3427080); Change from Baseline to Week 4; Test type: Superiority; p = 0.0002, Mixed-Effect Model Repeated Measures; Difference in LS means = -3.93, 95% CI 2-sided [-5.94 to -1.92]
Statistical Analysis 4: Comparison: Placebo vs 160 mg Elinzanetant (BAY3427080); Change from Baseline to Week 4; Test type: Superiority; p = 0.0115, Mixed-Effect Model Repeated Measures; Difference in LS means = -2.63, 95% CI 2-sided [-4.66 to -0.6]

2. Primary Outcome: Mean Change From Baseline in Mean Daily Frequency of Moderate and Severe Hot Flushes From Baseline to Week 12
Description: as for outcome 1
Time Frame: From baseline to Week 12
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot flushes per day
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Hot flushes per day
  Baseline | 11.82 (4.42) | 12.13 (8.81) | 14.55 (5.87) | 13.54 (7.17) | 12.92 (6.90)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 51 | 43
  Week 12: Change from baseline | -4.49 (4.29) | -6.48 (7.82) | -5.49 (5.31) | -7.91 (6.66) | -6.57 (5.83)
Statistical Analysis 1: Comparison: Placebo vs 40 mg Elinzanetant (BAY3427080); Change from Baseline to Week 12; Test type: Superiority; p = 0.2097, Mixed-Effect Model Repeated Measures; Difference in LS means = -1.67, 95% CI 2-sided [-4.28 to -0.95]
Statistical Analysis 2: Comparison: Placebo vs 80 mg Elinzanetant (BAY3427080); Change from Baseline to Week 12; Test type: Superiority; p = 0.6369, Mixed-Effect Model Repeated Measures; Difference in LS means = -0.77, 95% CI 2-sided [-3.97 to 2.44]
Statistical Analysis 3: Comparison: Placebo vs 120 mg Elinzanetant (BAY3427080); Change from Baseline to Week 12; Test type: Superiority; p = 0.0116, Mixed-Effect Model Repeated Measures; Difference in LS means = -2.95, 95% CI 2-sided [-5.22 to -0.67]
Statistical Analysis 4: Comparison: Placebo vs 160 mg Elinzanetant (BAY3427080); Change from Baseline to Week 12; Test type: Superiority; p = 0.1346, Mixed-Effect Model Repeated Measures; Difference in LS means = -1.78, 95% CI 2-sided [-4.12 to 0.56]

3. Primary Outcome: Mean Change From Baseline in Mean Severity of Moderate and Severe Hot Flushes From Baseline to Week 4
Description: Participants recorded daily in their eDiary the frequency and severity of hot flushes during the treatment period. Mean weekly severity = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). Severity is graded by the women from 1 to 3 (1 = mild; 2 = moderate; 3 = severe).
Time Frame: From baseline to Week 4
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot flushes per day
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Hot flushes per day
  Baseline | 2.54 (0.20) | 2.51 (0.26) | 2.63 (0.24) | 2.54 (0.24) | 2.54 (0.26)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 50 | 45
  Week 4: Change from baseline | -0.31 (0.41) | -0.38 (0.54) | -0.44 (0.56) | -0.51 (0.57) | -0.54 (0.67)
Statistical Analysis 1: Comparison: Placebo vs 40 mg Elinzanetant (BAY3427080); Change from Baseline to Week 4; Test type: Superiority; p = 0.7033, Mixed-Effect Model Repeated Measures; Difference in LS means = -0.05, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs 80 mg Elinzanetant (BAY3427080); Change from Baseline to Week 4; Test type: Superiority; p = 0.3724, Mixed-Effect Model Repeated Measures; Difference in LS means = -0.14, 95% CI 2-sided [-0.45 to 0.17]
Statistical Analysis 3: Comparison: Placebo vs 120 mg Elinzanetant (BAY3427080); Change from Baseline to Week 4; Test type: Superiority; p = 0.0896, Mixed-Effect Model Repeated Measures; Difference in LS means = -0.19, 95% CI 2-sided [-0.41 to 0.03]
Statistical Analysis 4: Comparison: Placebo vs 160 mg Elinzanetant (BAY3427080); Change from Baseline to Week 4; Test type: Superiority; p = 0.09, Mixed-Effect Model Repeated Measures; Difference in LS means = -0.19, 95% CI 2-sided [-0.41 to 0.03]

4. Primary Outcome: Mean Change From Baseline in Mean Severity of Moderate and Severe Hot Flushes From Baseline to Week 12
Description: Participants recorded daily in their eDiary the frequency and severity of hot flushes during the treatment period. Mean weekly severity = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). Severity was graded by the women from 1 to 3 (1 = mild; 2 = moderate; 3 = severe).
Time Frame: From baseline to Week 12
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot flushes per day
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Hot flushes per day
  Baseline | 2.54 (0.20) | 2.51 (0.26) | 2.63 (0.24) | 2.54 (0.24) | 2.54 (0.26)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 49 | 41
  Week 12: Change from baseline | -0.41 (0.50) | -0.53 (0.64) | -0.26 (0.45) | -0.56 (0.68) | -0.73 (0.78)
Statistical Analysis 1: Comparison: Placebo vs 40 mg Elinzanetant (BAY3427080); Change from Baseline to Week 12; Test type: Superiority; p = 0.5511, Mixed-Effect Model Repeated Measures; Difference in LS means = -0.09, 95% CI 2-sided [-0.39 to 0.21]
Statistical Analysis 2: Comparison: Placebo vs 80 mg Elinzanetant (BAY3427080); Change from Baseline to Week 12; Test type: Superiority; p = 0.3822, Mixed-Effect Model Repeated Measures; Difference in LS means = 0.16, 95% CI 2-sided [-0.2 to 0.52]
Statistical Analysis 3: Comparison: Placebo vs 120 mg Elinzanetant (BAY3427080); Change from Baseline to Week 12; Test type: Superiority; p = 0.2606, Mixed-Effect Model Repeated Measures; Difference in LS means = -0.15, 95% CI 2-sided [-0.41 to 0.11]
Statistical Analysis 4: Comparison: Placebo vs 160 mg Elinzanetant (BAY3427080); Change from Baseline to Week 12; Test type: Superiority; p = 0.0479, Mixed-Effect Model Repeated Measures; Difference in LS means = -0.27, 95% CI 2-sided [-0.53 to 0]

5. Secondary Outcome: Mean Change From Baseline in Frequency of Mean Daily Moderate and Severe Hot Flushes From Baseline to Weeks 1, 2, 8 and 16
Description: as for outcome 1
Time Frame: From baseline to Weeks 1, 2, 8 and 16
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot flushes per day
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Hot flushes per day
  Baseline | 11.82 (4.42) | 12.13 (8.81) | 14.55 (5.87) | 13.54 (7.17) | 12.92 (6.90)
  Week 1: Change from baseline | -1.22 (3.07) | -1.61 (3.05) | -1.63 (3.56) | -3.22 (3.43) | -3.09 (3.76)
  Week 2: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -2.19 (4.01) | -3.03 (3.95) | -3.47 (4.37) | -4.58 (4.70) | -3.78 (4.48)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 51 | 44
  Week 8: Change from baseline | -4.33 (4.79) | -5.72 (6.18) | -5.94 (5.26) | -7.84 (5.95) | -5.58 (6.00)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 42
  Week 16: Change from baseline | -3.95 (4.85) | -5.74 (9.45) | -2.01 (4.99) | -5.95 (6.95) | -2.78 (6.54)

6. Secondary Outcome: Mean Change From Baseline in Mean Severity of Moderate and Severe Hot Flushes From Baseline to Weeks 1, 2, 8 and 16
Description: Participants recorded daily in their diary the frequency and severity of hot flushes during the treatment period. Mean weekly severity = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). Severity is graded by the women from 1 to 3 (1 = mild; 2 = moderate; 3 = severe).
Time Frame: From baseline to Weeks 1, 2, 8 and 16
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot flushes per day
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 50 | 50
Hot flushes per day
  Baseline | 2.54 (0.20) | 2.51 (0.26) | 2.63 (0.24) | 2.54 (0.24) | 2.55 (0.26)
  Week 1: Change from baseline | -0.24 (0.30) | -0.21 (0.20) | -0.22 (0.21) | -0.25 (0.28) | -0.26 (0.26)
  Week 2: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 50 | 49
  Week 2: Change from baseline | -0.30 (0.39) | -0.32 (0.32) | -0.42 (0.58) | -0.37 (0.46) | -0.40 (0.55)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 50 | 42
  Week 8: Change from baseline | -0.45 (0.58) | -0.48 (0.54) | -0.40 (0.61) | -0.51 (0.54) | -0.65 (0.73)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 49 | 41
  Week 16: Change from baseline | 2.15 (0.65) | 2.03 (0.56) | 2.50 (0.46) | 2.13 (0.71) | 2.08 (0.62)

7. Secondary Outcome: Mean Change From Baseline in Mean Daily Frequency of All Hot Flushes From Baseline to Weeks 1, 2, 4, 8, 12 and 16
Description: as for outcome 1
Time Frame: From baseline to Weeks 1, 2, 4, 8, 12 and 16
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot flushes per day
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Hot flushes per day
  Baseline | 14.04 (5.57) | 14.19 (11.01) | 16.55 (6.89) | 15.39 (7.91) | 15.78 (9.62)
  Week 1 | -1.36 (3.03) | -1.72 (3.27) | -1.33 (5.68) | -3.30 (3.99) | -3.69 (4.81)
  Week 2: number analyzed (Participants) | 45 | 31 | 17 | 52 | 51
  Week 2 | -2.35 (4.60) | -2.99 (4.90) | -2.74 (5.97) | -4.57 (5.48) | -4.43 (5.68)
  Week 4: number analyzed (Participants) | 45 | 31 | 17 | 52 | 47
  Week 4 | -2.67 (4.09) | -4.11 (6.31) | -3.45 (8.54) | -6.70 (6.16) | -5.79 (6.09)
  Week 8: number analyzed (Participants) | 44 | 31 | 17 | 51 | 44
  Week 8 | -4.74 (5.57) | -5.65 (6.55) | -5.45 (6.56) | -7.96 (6.16) | -6.03 (6.43)
  Week 12: number analyzed (Participants) | 44 | 30 | 16 | 51 | 43
  Week 12 | -5.07 (5.48) | -6.50 (8.67) | -5.11 (8.41) | -7.94 (6.74) | -7.47 (7.13)
  Week 16: number analyzed (Participants) | 43 | 30 | 16 | 51 | 42
  Week 16 | -4.60 (6.17) | -5.83 (10.86) | -1.76 (7.50) | -6.19 (7.68) | -3.11 (6.71)

8. Secondary Outcome: Mean Change From Baseline in Mean Severity of All Hot Flushes From Baseline to Weeks 1, 2, 4, 8, 12 and 16
Description: as for outcome 6
Time Frame: From baseline to Weeks 1, 2, 4, 8, 12 and 16
Population: Participants with available data are reported.
Measure: Mean (Standard Deviation); unit: Hot flushes per day
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Hot flushes per day
  Baseline | 2.34 (0.32) | 2.34 (0.35) | 2.46 (0.37) | 2.38 (0.34) | 2.35 (0.39)
  Week 1: Change from baseline | -0.04 (0.23) | -0.04 (0.18) | -0.05 (0.12) | -0.09 (0.25) | -0.07 (0.18)
  Week 2: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -0.10 (0.32) | -0.15 (0.27) | -0.25 (0.52) | -0.21 (0.46) | -0.20 (0.50)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 52 | 47
  Week 4: Change from baseline | -0.11 (0.36) | -0.21 (0.47) | -0.27 (0.49) | -0.35 (0.60) | -0.34 (0.63)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 51 | 44
  Week 8: Change from baseline | -0.25 (0.54) | -0.31 (0.47) | -0.23 (0.52) | -0.35 (0.55) | -0.44 (0.72)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 51 | 43
  Week 12: Change from baseline | -0.21 (0.44) | -0.35 (0.57) | -0.08 (0.41) | -0.41 (0.62) | -0.52 (0.79)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 42
  Week 16: Change from baseline | -0.21 (0.49) | -0.30 (0.52) | 0.05 (0.34) | -0.26 (0.56) | -0.24 (0.54)

9. Secondary Outcome: Mean Change From Baseline in the Mean Daily Hot Flush Score (Frequency x Severity) at Weeks 1, 2, 4, 8, 12 and 16
Description: Mean daily Hot Flushes score = Sum of (frequency x severity) filled in the diary during the last 7 days (with at least one available data in the evening and/or morning) divided by 7. Severity is graded by the women from 1 to 3 (1 = mild; 2 = moderate; 3 = severe).
Time Frame: From baseline to Weeks 1, 2, 4, 8, 12 and 16
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: (units on a scale)*(hot flushes per day)
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
(units on a scale)*(hot flushes per day)
  Baseline | 32.35 (12.24) | 32.84 (24.82) | 40.76 (17.08) | 36.59 (19.88) | 35.73 (19.75)
  Week 1: Change from baseline | -3.09 (8.16) | -4.26 (7.93) | -4.18 (11.27) | -8.44 (8.98) | -8.67 (10.53)
  Week 2: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -5.62 (11.00) | -7.88 (10.77) | -9.08 (13.09) | -11.98 (12.39) | -10.51 (12.47)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 52 | 47
  Week 4: Change from baseline | -6.62 (9.79) | -10.68 (15.26) | -11.39 (18.82) | -17.54 (15.50) | -14.20 (14.30)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 51 | 44
  Week 8: Change from baseline | -11.63 (12.51) | -14.64 (16.33) | -16.17 (15.32) | -20.54 (15.80) | -14.89 (15.36)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 51 | 43
  Week 12: Change from baseline | -12.33 (11.96) | -16.71 (20.60) | -14.93 (16.83) | -20.72 (17.81) | -17.70 (15.38)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 42
  Week 16: Change from baseline | -10.89 (13.45) | -14.93 (25.48) | -4.97 (14.35) | -15.60 (19.03) | -7.50 (16.55)

10. Secondary Outcome: Number of Participants With ≥50% and ≥80% Reduction From Baseline in Mean Daily Hot Flushes Frequency at Week 12
Description: The percent change from baseline at a visit Week 12 was calculated. Percent change = (change from baseline in mean daily frequency of moderate and severe hot flushes from baseline to Week 12 / Mean daily frequency of moderate and severe hot flushes at baseline) * 100. A participant was considered as a responder with a reduction of ≥50% (or ≥80%) if the percent change was ≤-50 (or ≤-80).
Time Frame: Week 12
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 44 | 30 | 16 | 51 | 43
Participants
  >= 50% reduction: Yes | 17 | 20 | 5 | 32 | 30
  >= 50% reduction: No | 27 | 10 | 11 | 19 | 13
  >=80% reduction: Yes | 8 | 6 | 0 | 16 | 18
  >=80% reduction: No | 36 | 24 | 16 | 35 | 25

11. Secondary Outcome: Mean Change From Baseline in Number of All Night-time Awakenings (NTA) at Weeks 1, 2, 4, 8, 12 and 16
Description: Participants were provided with an eDiary to document the number of night-time awakenings (NTA). Each evening, participants recorded the total number of hot flushes of each severity experienced that day since waking. Each morning upon waking, subjects recorded the number of times they woke up in the night and the total number of hot flushes of each severity experienced during the night.
Time Frame: From baseline to Weeks 1, 2, 4, 8, 12 and 16
Population: Participants with available data are reported.
Measure: Mean (Standard Deviation); unit: Night-time awakenings per day
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Night-time awakenings per day
  Baseline | 3.86 (2.06) | 3.44 (1.82) | 5.00 (1.76) | 3.80 (2.20) | 3.85 (2.57)
  Week 1: Change from baseline | -0.65 (1.08) | -0.70 (1.24) | -0.57 (1.57) | -0.91 (1.06) | -0.86 (1.93)
  Week 2: Change from baseline: number analyzed (Participants) | 47 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -0.62 (1.54) | -0.70 (1.20) | -1.09 (1.84) | -1.10 (1.34) | -1.00 (2.10)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 52 | 47
  Week 4: Change from baseline | -0.86 (1.40) | -1.05 (1.43) | -0.99 (2.96) | -1.49 (1.43) | -1.03 (2.22)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 51 | 44
  Week 8: Change from baseline | -0.99 (1.31) | -1.66 (1.77) | -1.30 (2.15) | -1.79 (1.47) | -1.17 (2.51)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 51 | 43
  Week 12: Change from baseline | -1.28 (1.44) | -1.53 (1.89) | -1.61 (2.46) | -1.60 (1.38) | -1.40 (2.40)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 42
  Week 16: Change from baseline | -1.08 (1.30) | -0.96 (1.91) | -0.31 (2.90) | -1.05 (1.30) | -0.32 (2.10)

12. Secondary Outcome: Mean Change From Baseline in Mean Daily Number of NTAs Secondary to Hot Flushes at Weeks 1, 2, 4, 8, 12 and 16
Description: Subjects were provided with an eDiary to document the number of night-time awakenings (NTA). Each evening, subjects recorded the total number of hot flashes of each severity experienced that day since waking. Each morning upon waking, subjects recorded the number of times they woke up in the night and the total number of hot flushes of each severity experienced during the night. Night-time awakenings secondary to hot flashes corresponded to severe hot flash recorded on the morning diary, and all NTAs corresponded to the data recorded in the "Total number of times you woke up last night?" field from the eDiary recorded in the morning. Number of NTAs secondary to hot flushes could not be higher than the number of all NTAs.
Time Frame: From baseline to Weeks 1, 2, 4, 8, 12 and 16
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Night-time awakenings per day
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Night-time awakenings per day
  Baseline | 2.90 (1.64) | 2.41 (1.57) | 4.05 (1.86) | 2.76 (1.71) | 2.57 (1.54)
  Week 1: Change from baseline | -0.57 (0.96) | -0.52 (1.07) | -0.63 (1.53) | -0.90 (1.03) | -0.68 (1.14)
  Week 2: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -0.69 (1.03) | -0.75 (1.18) | -1.13 (1.89) | -1.18 (1.27) | -0.92 (1.38)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 52 | 47
  Week 4: Change from baseline | -0.89 (1.08) | -0.91 (1.26) | -1.33 (2.27) | -1.53 (1.19) | -1.01 (1.62)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 51 | 44
  Week 8: Change from baseline | -1.09 (1.36) | -1.50 (1.40) | -1.69 (2.21) | -1.79 (1.35) | -1.13 (1.86)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 51 | 43
  Week 12: Change from baseline | -1.31 (1.39) | -1.63 (1.46) | -1.70 (2.53) | -1.67 (1.27) | -1.32 (1.75)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 42
  Week 16: Change from baseline | -1.05 (1.19) | -1.29 (1.63) | -0.45 (2.05) | -1.19 (1.23) | -0.44 (1.62)

13. Secondary Outcome: Change From Baseline in the Global and Individual Domain Scores of the Pittsburgh Sleep Quality Index (PSQI) at Weeks 4, 8, 12 and 16
Description: The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. The PSQI uses 19 individual items to generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction, each scored 0 (no difficulty) to 3 (severe difficulty). The sum of scores for these seven components yields one global score (range 0 to 21). Higher scores indicated worse sleep quality.
Time Frame: From baseline to Weeks 4, 8, 12 and 16
Population: Participants in full analysis set (FAS) with evaluable data. Some participants either had missing value at baseline or missing value at a specific assessment week, so the change from baseline value cannot be obtained.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Units on scale
  Baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 50
  Baseline | 10.80 (2.39) | 11.94 (3.11) | 11.35 (3.66) | 10.80 (3.00) | 11.44 (3.14)
  Week 4: Change from baseline: number analyzed (Participants) | 41 | 31 | 17 | 50 | 45
  Week 4: Change from baseline | -0.63 (2.02) | -1.87 (2.93) | -1.94 (2.68) | -2.70 (3.11) | -2.80 (2.84)
  Week 8: Change from baseline: number analyzed (Participants) | 42 | 31 | 16 | 51 | 43
  Week 8: Change from baseline | -1.36 (2.90) | -2.39 (3.63) | -2.38 (3.30) | -3.00 (3.23) | -3.14 (3.37)
  Week 12: Change from baseline: number analyzed (Participants) | 41 | 30 | 16 | 49 | 41
  Week 12: Change from baseline | -1.15 (2.95) | -2.47 (3.82) | -2.81 (2.97) | -3.39 (3.12) | -3.54 (4.12)
  Week 16: Change from baseline: number analyzed (Participants) | 41 | 30 | 16 | 50 | 42
  Week 16: Change from baseline | -1.85 (2.46) | -2.10 (3.53) | -1.38 (3.26) | -2.24 (3.12) | -1.79 (2.69)

14. Secondary Outcome: Change From Baseline in the Insomnia Severity Index (ISI) Score at Weeks 4, 8, 12 and 16
Description: The ISI is a brief self-report questionnaire assessing the nature, severity, and impact of insomnia. The ISI comprises seven items assessing the perceived severity of difficulties initiating sleep, staying asleep, and early morning awakenings, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Participants rated each item on a scale of 0 to 4, yielding a total score ranging from 0 to 28.
  The total score was calculated by adding the scores for all seven items. Higher scores indicated severe insomnia.
Time Frame: From baseline to Weeks 4, 8, 12 and 16
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Units on scale
  Baseline: number analyzed (Participants) | 44 | 31 | 17 | 51 | 50
  Baseline | 12.43 (5.09) | 13.23 (5.36) | 13.24 (8.04) | 12.63 (5.66) | 13.74 (5.89)
  Week 4: Change from Baseline: number analyzed (Participants) | 40 | 31 | 17 | 50 | 45
  Week 4: Change from Baseline | -1.60 (2.98) | -2.74 (4.91) | -3.65 (6.03) | -5.14 (5.51) | -5.42 (5.42)
  Week 8: Change from Baseline: number analyzed (Participants) | 41 | 31 | 16 | 51 | 43
  Week 8: Change from Baseline | -1.51 (3.64) | -3.74 (5.63) | -4.44 (6.17) | -6.20 (4.93) | -5.72 (5.14)
  Week 12: Change from Baseline: number analyzed (Participants) | 40 | 30 | 16 | 49 | 41
  Week 12: Change from Baseline | -1.95 (4.70) | -3.80 (5.45) | -5.81 (5.86) | -6.12 (5.41) | -7.39 (5.82)
  Week 16: Change from Baseline: number analyzed (Participants) | 40 | 30 | 16 | 50 | 42
  Week 16: Change from Baseline | -2.65 (4.32) | -3.73 (6.02) | -3.00 (3.72) | -4.34 (5.58) | -4.00 (5.49)

15. Secondary Outcome: Change From Baseline in the Hot Flush Related Daily Interference Scale (HFRDIS) Scores at Weeks 2, 4, 8, 12 and 16
Description: The HFRDIS is a 10-item, self-report questionnaire assessing the impact of hot flushes on a woman's life during the past week. For each of the 10 items, participants rated how much hot flushes had interfered with that aspect of their life on a scale of 0 (not at all) to 10 (very much so). The total score was calculated by adding the scores for all 10 items. Higher scores indicated greater interference.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Units on scale
  Baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 50
  Baseline | 52.93 (18.40) | 52.74 (20.33) | 50.29 (21.45) | 53.86 (23.42) | 55.36 (19.71)
  Week 2: Change from baseline: number analyzed (Participants) | 42 | 31 | 17 | 51 | 48
  Week 2: Change from baseline | -4.00 (20.28) | -5.39 (21.99) | -11.12 (28.14) | -13.75 (29.66) | -10.90 (21.31)
  Week 4: Change from baseline: number analyzed (Participants) | 43 | 31 | 17 | 50 | 45
  Week 4: Change from baseline | -9.98 (20.84) | -13.00 (22.53) | -15.06 (24.02) | -23.04 (28.32) | -18.44 (23.37)
  Week 8: Change from baseline: number analyzed (Participants) | 42 | 31 | 16 | 51 | 43
  Week 8: Change from baseline | -15.48 (21.07) | -16.26 (23.71) | -17.88 (27.15) | -26.39 (24.90) | -24.09 (25.51)
  Week 12: Change from: number analyzed (Participants) | 41 | 30 | 16 | 49 | 41
  Week 12: Change from | -19.37 (20.20) | -21.30 (22.89) | -15.56 (28.70) | -28.33 (25.36) | -27.83 (24.64)
  Week 16: Change from baseline: number analyzed (Participants) | 41 | 30 | 16 | 50 | 42
  Week 16: Change from baseline | -15.22 (21.72) | -10.73 (24.87) | -16.69 (24.15) | -19.16 (22.43) | -12.07 (25.94)

16. Secondary Outcome: Change From Baseline in the Menopause-specific Quality-of-Life Questionnaire Intervention Version (MenQoL-I) Scores at Weeks 4, 8, 12 and 16
Description: The MenQoL-I is a validated questionnaire used to measure condition-specific quality of life in menopausal women. It is composed of 32 items across four domains (physical, vasomotor, psychosocial and sexual). For each item, participants recorded whether they had experienced the problem in the past month, and if so, they rated how bothered they were by the problem on a scale of 0 (not at all bothered) to 6 (extremely bothered). The item scores were converted to a score ranging from 1 to 8.
  Domain scores are calculated by averaging the converted individual item scores (range 1-8) related to the respective domain. (Domains: Vasomotor - items 1 to 3, Psychosocial - items 4 to 10, Physical- items 11- to 26, Sexual - items 27 to 29). For a MENQOL total score the aggregated mean of the mean domain scores is calculated. Higher scores indicate greater bother.
Time Frame: From baseline to Weeks 4, 8, 12 and 16;
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Units on scale
  Baseline: number analyzed (Participants) | 46 | 31 | 17 | 51 | 51
  Baseline | 4.00 (1.06) | 4.38 (1.16) | 4.47 (1.25) | 4.17 (1.13) | 4.50 (1.23)
  Week 4: Change from baseline: number analyzed (Participants) | 42 | 31 | 17 | 50 | 46
  Week 4: Change from baseline | -0.33 (0.90) | -0.62 (1.30) | -0.56 (0.87) | -1.29 (1.14) | -1.13 (1.09)
  Week 8: Change from baseline: number analyzed (Participants) | 43 | 31 | 16 | 51 | 43
  Week 8: Change from baseline | -0.62 (1.10) | -0.87 (1.25) | -0.91 (1.06) | -1.45 (1.18) | -1.50 (0.99)
  Week 12: Change from baseline: number analyzed (Participants) | 42 | 30 | 16 | 49 | 41
  Week 12: Change from baseline | -0.70 (1.03) | -0.81 (1.44) | -1.09 (0.76) | -1.54 (1.34) | -1.72 (1.32)
  Week 16: Change from baseline: number analyzed (Participants) | 42 | 30 | 16 | 50 | 42
  Week 16: Change from baseline | -0.68 (1.01) | -0.76 (1.33) | -0.69 (0.93) | -1.18 (1.13) | -1.00 (1.36)

17. Secondary Outcome: Change From Baseline in the Beck Depression Inventory II (BDI-II) Scores at Weeks 2, 4, 8, 12 and 16
Description: The BDI-II is a 21-item questionnaire assessing the intensity of depressive symptoms over the past 2 weeks. It is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex. Participants rated each item on a scale of 0 to 3 to give a total score ranging from 0 to 63, with a higher score suggesting more severe depressive symptoms.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Units on scale
  Baseline: number analyzed (Participants) | 44 | 31 | 17 | 51 | 50
  Baseline | 11.18 (8.74) | 14.29 (11.36) | 10.47 (7.01) | 9.92 (8.62) | 11.48 (9.30)
  Week 2: Change from baseline: number analyzed (Participants) | 41 | 31 | 17 | 51 | 48
  Week 2: Change from baseline | -1.90 (5.29) | -2.23 (9.27) | -3.06 (7.34) | -3.65 (6.95) | -2.71 (6.08)
  Week 4: Change from baseline: number analyzed (Participants) | 42 | 31 | 17 | 50 | 45
  Week 4: Change from baseline | -1.55 (5.14) | -4.23 (9.82) | -2.35 (5.16) | -4.08 (6.39) | -4.13 (6.63)
  Week 8: Change from baseline: number analyzed (Participants) | 41 | 31 | 16 | 51 | 43
  Week 8: Change from baseline | -2.24 (5.26) | -5.32 (10.13) | -2.00 (8.22) | -4.73 (6.34) | -5.51 (7.14)
  Week 12: Change from baseline: number analyzed (Participants) | 40 | 30 | 16 | 49 | 41
  Week 12: Change from baseline | -1.30 (7.22) | -5.00 (3.80) | -1.69 (7.65) | -4.29 (6.56) | -5.73 (7.39)
  Week 16: Change from baseline: number analyzed (Participants) | 40 | 30 | 16 | 50 | 42
  Week 16: Change from baseline | -2.43 (6.08) | -5.10 (11.62) | -0.75 (6.71) | -4.04 (6.12) | -2.36 (8.05)

18. Secondary Outcome: Plasma Elinzanetant Concentrations at Weeks 2, 4, 8 ,12
Description: Blood samples for analysis of plasma elinzanetant concentrations were collected at Weeks 2, 4, 8, and 12. A small number of participants had elinzanetant concentrations below the LOQ for the assay (1.5 ng/mL) at two or more visits (three participants in each of the 40 mg, 120 mg, and 160 mg groups, four in 80 mg group), indicating that these subjects were non compliant with treatment.
Time Frame: At Weeks 2, 4, 8 ,12
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 31 | 17 | 52 | 52
ng/ml
  Week 2 | 64.254 (75.681) [lower limit 75.681] | 157.207 (93.120) [lower limit 93.120] | 292.929 (100.381) [lower limit 100.381] | 319.552 (170.571) [lower limit 170.571]
  Week 4 | 78.946 (78.892) [lower limit 78.892] | 118.554 (175.865) [lower limit 175.865] | 253.800 (142.944) [lower limit 142.944] | 398.389 (91.644) [lower limit 91.644]
  Week 8 | 87.985 (68.277) [lower limit 68.277] | 138.795 (72.619) [lower limit 72.619] | 226.121 (79.171) [lower limit 79.171] | 341.673 (145.535) [lower limit 145.535]
  Week 12 | 70.138 (66.542) [lower limit 66.542] | 130.729 (414.199) [lower limit 414.199] | 197.041 (231.390) [lower limit 231.390] | 298.896 (220.963) [lower limit 220.963]

19. Secondary Outcome: Nature and Severity of Adverse Events
Description: A Treatment-Emergent Adverse Events (TEAE) is defined as any adverse event (serious and non-serious) with the onset date on or after the date of first dosing with study treatment. Safety Analysis Set.
Time Frame: Up to Week 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Participants
  Number of TEAEs | 28 | 17 | 14 | 34 | 38
  Number of TEAEs related to IMP | 7 | 7 | 8 | 8 | 12
  Number of Serious TEAEs | 2 | 0 | 1 | 1 | 1
  Number of TEAEs leading to death | 0 | 0 | 0 | 0 | 0
  Number of Severe TEAEs | 2 | 0 | 1 | 3 | 2

20. Secondary Outcome: Withdrawals Due to an Adverse Event
Description: A Treatment-Emergent Adverse Events (TEAE) is defined as any adverse event (serious and non-serious) with the onset date on or after the date of first dosing with study treatment.
Time Frame: Up to Week 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Participants
  TEAEs leading to treatment discontinuation | 1 | 0 | 2 | 0 | 5
  TEAEs leading to study discontinuation | 1 | 0 | 1 | 0 | 4

21. Secondary Outcome: Number of Subjects Used Concomitant Medications
Description: A concomitant medication is defined as any medication used on or after date and time of first randomised treatment. All concomitant medications taken during the study were recorded in the eCRF. Any medication that was not specifically prohibited was allowed. (1) Antidiarrheals, intestinal antiinflammatory/antiinfective agents.
Time Frame: Up to Week 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Participants
  Analgesics | 18 | 8 | 9 | 12 | 16
  Antiinflammatory and antirheumatic products | 14 | 7 | 5 | 12 | 13
  Vitamins | 14 | 6 | 6 | 9 | 14
  Drugs for acid related disorders | 13 | 7 | 2 | 10 | 10
  Psychoanaleptics | 6 | 5 | 4 | 10 | 9
  Psycholeptics | 3 | 7 | 5 | 7 | 7
  Antibacterials for systemic use | 9 | 5 | 2 | 5 | 7
  Drugs for obstructive airway diseases | 7 | 3 | 3 | 4 | 9
  Lipid modifying agents | 3 | 3 | 4 | 8 | 4
  Agents acting on the renin-angiotensin system | 7 | 4 | 0 | 11 | 3
  Thyroid therapy | 4 | 3 | 3 | 7 | 5
  Antihistamines for systemic use | 5 | 4 | 3 | 6 | 3
  Antithrombotic agents | 2 | 4 | 2 | 6 | 4
  Nasal preparations | 2 | 4 | 1 | 1 | 7
  Diuretics | 1 | 2 | 0 | 5 | 5
  Antianemic preparations | 5 | 2 | 2 | 5 | 2
  Mineral supplements | 2 | 2 | 3 | 3 | 3
  Calcium channel blockers | 3 | 0 | 1 | 6 | 3
  Drugs used in diabetes | 3 | 2 | 0 | 1 | 6
  Beta blocking agents | 1 | 2 | 0 | 5 | 1
  Ophthalmologicals | 1 | 1 | 2 | 3 | 1
  Urologicals | 1 | 1 | 1 | 3 | 1
  Antidiarrheals, intestinal agents (1) | 2 | 2 | 0 | 0 | 3
  Antivirals for systemic use | 1 | 3 | 1 | 1 | 0
  Corticosteroids for systemic use | 1 | 1 | 0 | 1 | 3
  Drugs for constipation | 2 | 0 | 1 | 3 | 1
  Anesthetics | 2 | 1 | 0 | 3 | 0
  Antiemetics and antinauseants | 2 | 0 | 1 | 1 | 2
  Drugs for functional gastrointestinal disorders | 3 | 1 | 0 | 1 | 2
  General nutrients | 1 | 1 | 0 | 1 | 2
  Topical products for joint and muscular pain | 1 | 2 | 0 | 0 | 2
  Antifungals for dermatological use | 0 | 1 | 1 | 0 | 1
  Antiobesity preparations, excl. Diet products | 0 | 0 | 0 | 2 | 1
  Corticosteroids, dermatological preparations | 1 | 2 | 0 | 1 | 0
  Cough and cold preparations | 3 | 1 | 0 | 2 | 0
  Other nervous system drugs | 1 | 1 | 0 | 1 | 1
  Unspecified herbal and traditional medicine | 1 | 0 | 1 | 1 | 1
  All other therapeutic products | 0 | 0 | 0 | 1 | 0
  Anti-acne preparations | 0 | 1 | 0 | 1 | 0
  Other alimentary tract and metabolism products | 1 | 1 | 0 | 1 | 0
  Throat preparations | 0 | 1 | 0 | 0 | 1
  Vaccines | 0 | 1 | 0 | 1 | 0
  Antiepileptics | 0 | 0 | 1 | 0 | 0
  Antihemorrhagics | 0 | 0 | 0 | 0 | 1
  Antihypertensives | 0 | 0 | 1 | 0 | 0
  Antiprotozoals | 0 | 0 | 0 | 0 | 1
  Antipruritics, incl. antihistamines, anesthetics | 0 | 0 | 0 | 0 | 1
  Antipsoriatics | 0 | 0 | 0 | 0 | 1
  Bile and liver therapy | 0 | 0 | 0 | 1 | 0
  Drugs for treatment of bone diseases | 0 | 0 | 1 | 0 | 0
  Gynecological antiinfectives and antiseptics | 0 | 0 | 0 | 1 | 0
  Immunosuppressants | 0 | 0 | 0 | 1 | 0
  Other respiratory system products | 0 | 0 | 0 | 0 | 1
  Stomatological preparations | 0 | 0 | 0 | 0 | 1
  Tonics | 0 | 0 | 0 | 1 | 0
  Muscle relaxants | 2 | 0 | 1 | 1 | 2
  Antibiotics,chemotherapeutics (dermatological use) | 1 | 0 | 0 | 1 | 0
  Antimycotics for systemic use | 1 | 0 | 0 | 0 | 0

22. Secondary Outcome: Change From Baseline in Vital Signs (Systolic Blood Pressure) at Weeks 2, 4, 8, 12 and 16
Description: Vital signs, including systolic and diastolic blood pressure, pulse rate, temperature, weight, waist circumference, and height, were measured at the time points and recorded in the eCRF. All vital signs were reviewed by the Investigator or delegated physician.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
mmHg
  Baseline | 123.2 (10.4) | 124.2 (10.1) | 128.9 (9.8) | 124.6 (10.9) | 124.0 (12.9)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | 0.3 (12.5) | -0.2 (9.0) | -1.5 (12.5) | -2.9 (9.3) | -0.8 (9.2)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | 1.7 (12.4) | 0.1 (11.9) | -3.1 (9.4) | -4.7 (10.7) | -1.3 (10.8)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 16 | 52 | 46
  Week 8: Change from baseline | 0.5 (10.8) | 0.5 (12.5) | -2.1 (10.1) | -1.3 (10.0) | -3.8 (10.5)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | -0.6 (12.2) | -2.1 (10.9) | -5.9 (11.3) | -1.1 (10.2) | -1.3 (12.8)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | 3.8 (13.3) | -0.9 (11.7) | -6.4 (11.1) | -1.4 (10.8) | 2.1 (9.4)

23. Secondary Outcome: Change From Baseline in Vital Signs (Diastolic Blood Pressure) at Weeks 2, 4, 8, 12 and 16
Description: Vital signs, including systolic and diastolic blood pressure were measured at the time points and recorded in the eCRF. All vital signs were reviewed by the Investigator or delegated physician.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
mmHg
  Baseline | 80.1 (8.0) | 78.7 (8.5) | 79.9 (9.1) | 78.1 (7.6) | 78.7 (10.1)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 16 | 52 | 51
  Week 2: Change from baseline | -0.7 (6.6) | -1.1 (8.4) | -0.8 (8.7) | -3.1 (7.6) | -0.4 (7.6)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | -0.2 (7.4) | 1.2 (7.8) | -2.1 (6.5) | -2.8 (9.1) | -2.3 (8.0)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 16 | 52 | 46
  Week 8: Change from baseline | 0.2 (6.7) | -0.5 (6.8) | -3.6 (6.9) | -0.6 (8.4) | -1.6 (7.5)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | -0.5 (9.6) | -2.8 (9.9) | -2.2 (7.1) | -1.8 (10.3) | -1.0 (9.3)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | 1.6 (7.6) | -1.2 (8.3) | -3.8 (9.7) | -1.9 (9.1) | 0.6 (7.2)

24. Secondary Outcome: Change From Baseline in Vital Signs (Pulse Rate) at Weeks 2, 4, 8, 12 and 16
Description: as for outcome 22
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
beats/min
  Baseline | 69.7 (7.8) | 71.4 (10.3) | 70.6 (8.7) | 70.1 (10.2) | 69.7 (10.2)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -0.1 (8.1) | -0.3 (7.3) | -0.7 (9.9) | -3.1 (9.7) | 2.1 (9.4)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | -0.6 (6.9) | 0.5 (7.6) | -2.8 (8.9) | -1.8 (6.4) | 0.9 (7.7)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 16 | 52 | 46
  Week 8: Change from baseline | 0.4 (7.7) | -0.5 (8.1) | -3.1 (9.8) | -2.8 (7.9) | 0.3 (8.1)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | 0.1 (9.2) | 0.3 (8.4) | 0.9 (8.8) | -1.4 (8.8) | 0.9 (7.4)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | 3.2 (10.6) | 3.3 (10.5) | 0.0 (11.3) | -0.7 (8.5) | 0.3 (8.4)

25. Secondary Outcome: Change From Baseline in Vital Signs (Temperature) at Weeks 2, 4, 8, 12 and 16
Description: as for outcome 22
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: Celsius (C)
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Celsius (C)
  Baseline | 36.69 (0.43) | 36.62 (0.32) | 36.73 (0.30) | 36.52 (0.46) | 36.68 (0.39)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -0.09 (0.40) | -0.04 (0.28) | 0.04 (0.26) | 0.12 (0.50) | -0.01 (0.43)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 50 | 48
  Week 4: Change from baseline | -0.15 (0.47) | -0.06 (0.34) | 0.01 (0.41) | 0.12 (0.46) | -0.06 (0.32)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 16 | 52 | 46
  Week 8: Change from baseline | -0.09 (0.38) | -0.01 (0.35) | 0.00 (0.31) | 0.11 (0.49) | -0.01 (0.42)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | -0.12 (0.44) | -0.12 (0.31) | -0.03 (0.38) | 0.04 (0.46) | -0.08 (0.36)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | -0.07 (0.50) | -0.03 (0.30) | -0.04 (0.32) | 0.08 (0.41) | -0.09 (0.41)

26. Secondary Outcome: Change From Baseline in Vital Signs (Weight) at Weeks 2, 4, 8, 12 and 16
Description: as for outcome 22
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Kilogram (Kg)
  Baseline | 75.85 (13.13) | 72.65 (14.76) | 78.14 (15.75) | 72.36 (15.26) | 74.11 (15.02)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | 0.20 (1.07) | 0.30 (1.03) | 0.13 (1.32) | -0.13 (1.19) | 0.04 (0.84)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | 0.23 (1.51) | 0.08 (1.11) | 0.12 (1.88) | -0.31 (1.26) | 0.00 (1.35)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 16 | 52 | 46
  Week 8: Change from baseline | 0.16 (1.98) | 0.26 (1.59) | -0.11 (1.79) | -0.18 (1.78) | -0.25 (2.32)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | -0.02 (2.34) | 0.58 (2.46) | -0.14 (2.03) | -0.08 (1.93) | -0.48 (2.62)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | 0.17 (2.48) | 0.39 (2.81) | -0.13 (2.59) | -0.20 (2.13) | -0.34 (2.82)

27. Secondary Outcome: Change From Baseline in Vital Signs (Body Mass Index ) at Weeks 2, 4, 8, 12 and 16
Description: as for outcome 22
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
kg/m^2
  Baseline | 28.59 (3.81) | 27.69 (4.97) | 29.81 (4.93) | 27.26 (4.85) | 27.72 (4.74)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | 0.07 (0.41) | 0.11 (0.39) | 0.06 (0.5) | -0.04 (0.45) | 0.01 (0.33)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | 0.07 (0.58) | 0.02 (0.42) | 0.06 (0.75) | -0.11 (0.49) | 0.00 (0.53)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 16 | 52 | 46
  Week 8: Change from baseline | 0.04 (0.75) | 0.09 (0.59) | -0.04 (0.69) | -0.06 (0.66) | -0.09 (0.88)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | -0.03 (0.87) | 0.21 (0.87) | -0.05 (0.79) | -0.02 (0.73) | -0.18 (0.99)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | 0.04 (0.96) | 0.13 (1.01) | -0.04 (1.01) | -0.07 (0.79) | -0.13 (1.07)

28. Secondary Outcome: Change From Baseline in Vital Signs (Waist Circumference) at Weeks 2, 4, 8, 12 and 16
Description: as for outcome 22
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
cm
  Baseline: number analyzed (Participants) | 46 | 31 | 17 | 50 | 52
  Baseline | 95.47 (11.69) | 93.61 (13.10) | 97.59 (13.15) | 91.12 (13.03) | 92.42 (12.36)
  Week 2: Change from baseline: number analyzed (Participants) | 43 | 31 | 17 | 49 | 51
  Week 2: Change from baseline | 0.26 (3.99) | 0.79 (3.55) | -0.91 (2.15) | 0.13 (3.72) | -0.18 (3.90)
  Week 4: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 48 | 48
  Week 4: Change from baseline | 0.17 (4.99) | -0.07 (4.23) | -1.26 (3.00) | 0.05 (3.84) | -0.09 (3.97)
  Week 8: Change from baseline: number analyzed (Participants) | 43 | 31 | 16 | 50 | 45
  Week 8: Change from baseline | -0.14 (4.45) | -0.11 (4.30) | 0.04 (2.77) | -0.76 (4.10) | -0.08 (4.71)
  Week 12: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 48 | 45
  Week 12: Change from baseline | -1.72 (5.25) | -1.16 (4.87) | 0.60 (2.81) | -0.25 (3.97) | -0.39 (4.42)
  Week 16: Change from baseline: number analyzed (Participants) | 42 | 30 | 16 | 49 | 44
  Week 16: Change from baseline | -0.80 (5.46) | -0.99 (5.18) | 4.33 (12.90) | 0.02 (4.58) | -0.24 (4.41)

29. Secondary Outcome: Number of Subjects With Normal Electrocardiogram (ECG) Findings at Each Visit
Description: All ECGs were performed after the subject had rested for 5 minutes in a semi-recumbent position. All ECG reports were reviewed, signed and dated by the Investigator or delegated physician. Reported results are cardiovascular system-examination findings. Normal ECG was decided by investigator. The findings are presented as Normal ECG.
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Participants
  Baseline | 38 | 24 | 11 | 31 | 34
  Week 2: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 | 33 | 23 | 12 | 34 | 27
  Week 4: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 | 32 | 23 | 10 | 28 | 31
  Week 8: number analyzed (Participants) | 44 | 31 | 17 | 52 | 46
  Week 8 | 29 | 21 | 12 | 30 | 27
  Week 12: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12 | 30 | 22 | 11 | 31 | 31
  Week 16: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16 | 27 | 26 | 14 | 31 | 28

30. Secondary Outcome: Number of Subjects With Abnormal Not Clinically Significant ECG Findings at Each Visit
Description: All ECGs were performed after the subject had rested for 5 minutes in a semi-recumbent position. All ECG reports were reviewed, signed and dated by the Investigator or delegated physician. Reported results are cardiovascular system-examination findings. Abnormal not clinically significant ECG findings were decided by investigator. The findings are presented as Abnormal not clinically significant ECG.
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Participants
  Baseline | 9 | 7 | 6 | 21 | 18
  Week 2: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 | 11 | 8 | 5 | 18 | 24
  Week 4: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 | 13 | 8 | 6 | 23 | 17
  Week 8: number analyzed (Participants) | 44 | 31 | 17 | 52 | 46
  Week 8 | 15 | 10 | 5 | 21 | 19
  Week 12: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12 | 14 | 8 | 5 | 19 | 14
  Week 16: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16 | 16 | 4 | 2 | 20 | 17

31. Secondary Outcome: Number of Subjects With Abnormal Clinically Significant ECG Findings at Each Visit
Description: All ECGs were performed after the subject had rested for 5 minutes in a semi-recumbent position. All ECG reports were reviewed, signed and dated by the Investigator or delegated physician. Reported results are cardiovascular system-examination findings. Abnormal clinically significant ECG findings were decided by investigator. The findings are presented as Abnormal clinically significant ECG.
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Participants
  Baseline | 0 | 0 | 0 | 0 | 0
  Week 2: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 | 0 | 0 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 | 0 | 0 | 1 | 0 | 0
  Week 8: number analyzed (Participants) | 44 | 31 | 17 | 52 | 46
  Week 8 | 0 | 0 | 0 | 1 | 0
  Week 12: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12 | 0 | 0 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Change From Baseline at Weeks 2, 4, 8, 12 and 16 in ECG Intervals (RR)
Description: All ECGs were performed after the subject had rested for 5 minutes in a semi-recumbent position. The same model of ECG recorder was used throughout the study for any given subject wherever possible. All ECG reports were reviewed, signed and dated by the Investigator or delegated physician. Reports were then filed with the subject's medical record. In categories the number of subjects analyzed (N) for each week is mentioned for each reporting group respectively.
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: mSec
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
mSec
  Baseline | 913.5 (128.5) | 891.4 (145.6) | 934.3 (120.3) | 927.8 (135.5) | 935.9 (151.2)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | 17.3 (84.2) | 23.0 (101.7) | -12.6 (99.7) | 27.3 (94.7) | -2.6 (137.7)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | 1.6 (82.8) | 24.8 (101.9) | 20.5 (108.5) | 27.3 (92.6) | 4.5 (108.0)
  Week 8: Change from baseline ): number analyzed (Participants) | 44 | 31 | 17 | 52 | 46
  Week 8: Change from baseline ) | 35.8 (108.7) | 24.8 (104.6) | 19.0 (128.6) | 22.3 (109.2) | -22.6 (90.1)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | 25.5 (143.4) | 18.0 (110.9) | -23.3 (105.1) | 27.2 (95.9) | -1.4 (107.9)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | -22.4 (135.5) | 2.4 (138.5) | -25.4 (149.6) | 5.9 (110.8) | -8.0 (110.3)

33. Secondary Outcome: Change From Baseline at Weeks 2, 4, 8, 12 and 16 in ECG Intervals (PR)
Description: All ECGs were performed after the subject had rested for 5 minutes in a semi-recumbent position. The same model of ECG recorder was used throughout the study for any given subject wherever possible. All ECG reports were reviewed, signed and dated by the Investigator or delegated physician. Reports were then filed with the subject's medical record.
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: mSec
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
mSec
  Baseline | 162.6 (21.8) | 167.8 (16.5) | 162.9 (21.7) | 157.2 (21.7) | 164.2 (25.8)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | 1.2 (9.7) | 4.6 (11.7) | 5.2 (11.8) | 3.0 (10.2) | -2.2 (16.3)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | 0.0 (11.2) | 5.9 (12.3) | 2.9 (12.1) | 3.8 (17.7) | 1.8 (13.8)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 46
  Week 8: Change from baseline | 1.5 (15.1) | 3.6 (10.4) | -0.1 (12.3) | 4.3 (10.3) | -1.1 (14.5)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | 1.6 (11.5) | 3.9 (11.7) | 0.7 (16.2) | 1.9 (11.4) | -1.5 (16.9)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | 0.4 (11.3) | 2.2 (13.3) | 2.4 (16.0) | 2.8 (11.1) | -0.4 (13.3)

34. Secondary Outcome: Change From Baseline at Weeks 2, 4, 8, 12 and 16 in ECG Intervals (QT)
Description: as for outcome 33
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: mSec
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
mSec
  Baseline | 394.5 (31.2) | 397.2 (28.7) | 403.5 (26.9) | 402.3 (40.3) | 401.2 (28.0)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | 3.6 (18.0) | 0.2 (17.8) | 1.1 (21.7) | -0.9 (35.6) | -3.2 (25.2)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | 4.7 (18.5) | -0.1 (18.5) | 4.8 (35.2) | 0.2 (28.1) | 0.8 (21.5)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 46
  Week 8: Change from baseline | 2.0 (19.0) | 1.5 (17.2) | 6.5 (28.4) | 0.5 (34.6) | -4.0 (20.3)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | 1.4 (25.1) | 0.8 (21.6) | -8.9 (20.6) | -1.1 (32.9) | 1.0 (19.5)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | -1.7 (23.3) | -4.7 (24.4) | -3.2 (27.6) | -4.1 (38.1) | -2.4 (25.5)

35. Secondary Outcome: Change From Baseline at Weeks 2, 4, 8, 12 and 16 in ECG Intervals (QTc)
Description: All ECGs were performed after the subject had rested for 5 minutes in a semi-recumbent position. The same model of ECG recorder was used throughout the study for any given subject wherever possible. All ECG reports were reviewed, signed and dated by the Investigator or delegated physician. Reports were then filed with the subject's medical record. QTc: QT corrected interval.
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: mSec
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
mSec
  Baseline | 410.6 (20.9) | 417.9 (21.4) | 416.4 (14.1) | 415.9 (29.3) | 415.2 (22.1)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | 1.6 (14.3) | -2.4 (11.2) | 2.9 (14.7) | -4.9 (28.2) | -2.1 (15.4)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | 5.6 (16.1) | -5.4 (11.8) | 1.7 (19.9) | -2.9 (24.5) | 0.2 (16.3)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 46
  Week 8: Change from baseline | -3.9 (18.5) | -3.8 (12.3) | 2.3 (10.8) | -2.2 (27.5) | 1.2 (14.7)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | -2.4 (20.8) | -3.2 (14.9) | -3.1 (14.4) | -4.7 (31.3) | 0.5 (14.4)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | 2.8 (14.9) | -4.8 (13.6) | 4.3 (17.5) | -4.5 (31.2) | -1.6 (13.6)

36. Secondary Outcome: Change From Baseline at Weeks 2, 4, 8, 12 and 16 in ECG Intervals (QTcF)
Description: All ECGs were performed after the subject had rested for 5 minutes in a semi-recumbent position. The same model of ECG recorder was used throughout the study for any given subject wherever possible. All ECG reports were reviewed, signed and dated by the Investigator or delegated physician. Reports were then filed with the subject's medical record. QTcF: QT interval with Fridericia's correction.
Time Frame: At Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: mSec
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
mSec
  Baseline | 407.2 (20.6) | 413.8 (19.9) | 413.2 (14.3) | 413.1 (30.7) | 411.4 (18.6)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | 1.2 (13.7) | -3.5 (10.2) | 3.4 (13.4) | -4.8 (29.5) | -2.5 (15.7)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | 4.8 (16.4) | -4.2 (11.5) | 2.1 (23.4) | -3.5 (24.7) | 0.4 (15.4)
  Week 8: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 46
  Week 8: Change from baseline | -2.8 (15.9) | -2.7 (10.9) | 4.0 (13.2) | -2.6 (28.7) | -0.4 (16.1)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 45
  Week 12: Change from baseline | -1.7 (18.5) | -1.9 (13.9) | -5.1 (13.2) | -5.1 (30.8) | 1.1 (14.6)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | 2.6 (15.1) | -5.6 (14.2) | 1.5 (14.5) | -4.8 (32.7) | -1.3 (16.4)

37. Secondary Outcome: Number of Subjects With Absolute QTcF Values by Category at Each Visit: ≤450, >450 to ≤480, >480 to ≤500, >500 Msec
Description: Absolute QTcF values reported.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Participants
  Baseline: missing | 0 | 0 | 0 | 0 | 0
  Baseline: <=450 msec | 46 | 30 | 16 | 51 | 50
  Baseline: >450 to <=480 msec | 1 | 1 | 1 | 0 | 2
  Baseline: >480 to <=500 msec | 0 | 0 | 0 | 0 | 0
  Baseline: >500 msec | 0 | 0 | 0 | 1 | 0
  Week 2: missing | 3 | 0 | 0 | 0 | 1
  Week 2: <=450 msec | 44 | 30 | 16 | 52 | 50
  Week 2: >450 to <=480 msec | 0 | 1 | 1 | 0 | 1
  Week 2: >480 to <=500 msec | 0 | 0 | 0 | 0 | 0
  Week 2: >500 msec | 0 | 0 | 0 | 0 | 0
  Week 4: missing | 2 | 0 | 0 | 1 | 4
  Week 4: <=450 msec | 44 | 30 | 16 | 51 | 47
  Week 4: >450 to <=480 msec | 1 | 1 | 0 | 0 | 1
  Week 4: >480 to <=500 msec | 0 | 0 | 0 | 0 | 0
  Week 4: >500 msec | 0 | 0 | 1 | 0 | 0
  Week 8: missing | 3 | 0 | 0 | 0 | 6
  Week 8: <=450 msec | 44 | 30 | 17 | 52 | 46
  Week 8: >450 to <=480 msec | 0 | 1 | 0 | 0 | 0
  Week 8: >480 to <=500 msec | 0 | 0 | 0 | 0 | 0
  Week 8: >500 msec | 0 | 0 | 0 | 0 | 0
  Week 12: missing | 3 | 1 | 1 | 2 | 7
  Week 12: <=450 msec | 44 | 30 | 16 | 50 | 45
  Week 12: >450 to <=480 msec | 0 | 0 | 0 | 0 | 0
  Week 12: >480 to <=500 msec | 0 | 0 | 0 | 0 | 0
  Week 12: >500 msec | 0 | 0 | 0 | 0 | 0
  Week 16: missing | 4 | 1 | 1 | 1 | 7
  Week 16: <=450 msec | 42 | 30 | 15 | 51 | 44
  Week 16: >450 to <=480 msec | 1 | 0 | 1 | 0 | 1
  Week 16: >480 to <=500 msec | 0 | 0 | 0 | 0 | 0
  Week 16: >500 msec | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: Number of Subjects With Change From Baseline in ECG QTcF Values by Category at Weeks 2, 4, 8, 12 and 16: ≤0, >0 to ≤30, >30 to ≤60, >60 Msec
Description: Increase from Baseline overtime was reported.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Participants
  Week 2: missing | 3 | 0 | 0 | 0 | 1
  Week 2: <=0 msec | 19 | 21 | 8 | 27 | 29
  Week 2: >0 to <=30 msec | 25 | 10 | 8 | 24 | 22
  Week 2: >30 to <=60 msec | 0 | 0 | 1 | 1 | 0
  Week 2: >60 msec | 0 | 0 | 0 | 0 | 0
  Week 4: missing | 2 | 0 | 0 | 1 | 4
  Week 4: <=0 msec | 20 | 20 | 8 | 27 | 24
  Week 4: >0 to <=30 msec | 23 | 11 | 8 | 24 | 22
  Week 4: >30 to <=60 msec | 2 | 0 | 0 | 0 | 2
  Week 4: >60 msec | 0 | 0 | 1 | 0 | 0
  Week 8: missing | 3 | 0 | 0 | 0 | 6
  Week 8: <=0 msec | 24 | 20 | 8 | 25 | 19
  Week 8: >0 to <=30 msec | 20 | 11 | 9 | 26 | 26
  Week 8: >30 to <=60 msec | 0 | 0 | 0 | 1 | 1
  Week 8: >60 msec | 0 | 0 | 0 | 0 | 0
  Week 12: missing | 3 | 1 | 1 | 2 | 7
  Week 12: <=0 msec | 24 | 15 | 10 | 29 | 22
  Week 12: >0 to <=30 msec | 19 | 15 | 6 | 21 | 22
  Week 12: >30 to <=60 msec | 1 | 0 | 0 | 0 | 1
  Week 12: >60 msec | 0 | 0 | 0 | 0 | 0
  Week 16: missing | 4 | 1 | 1 | 1 | 7
  Week 16: <=0 msec | 18 | 18 | 7 | 26 | 24
  Week 16: >0 to <=30 msec | 23 | 12 | 9 | 24 | 20
  Week 16: >30 to <=60 msec | 2 | 0 | 0 | 1 | 1
  Week 16: >60 msec | 0 | 0 | 0 | 0 | 0

39. Secondary Outcome: Change From Baseline in the Electronic Columbia Suicide Severity Rating Scale (eC-SSRS) at Weeks 4, 12 and 16
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) is a rating scale created to evaluate suicidality in adults and children over the age of 12. It rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The version used was the eC-SSRS, which is a subject-reported version of the scale. Shifts from baseline versus post-baseline to demonstrate changes in categories (cat) were reported using cat 1 (No Suicidal Ideation or Behaviour), cat 2 (Suicidal Ideation) and cat 3 (Suicidal Behaviour).
Time Frame: Baseline to Weeks 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 42 | 27 | 16 | 46 | 46
Participants
  Week 4: shift from cat 1 to cat 1: number analyzed (Participants) | 42 | 26 | 16 | 44 | 46
  Week 4: shift from cat 1 to cat 1 | 34 | 14 | 13 | 38 | 38
  Week 4: shift from cat 1 to cat 2: number analyzed (Participants) | 42 | 26 | 16 | 44 | 46
  Week 4: shift from cat 1 to cat 2 | 1 | 0 | 0 | 0 | 0
  Week 4: shift from cat 1 to cat 3: number analyzed (Participants) | 42 | 26 | 16 | 44 | 46
  Week 4: shift from cat 1 to cat 3 | 0 | 0 | 0 | 0 | 0
  Week 4: shift from cat 2 to cat 1: number analyzed (Participants) | 42 | 26 | 16 | 44 | 46
  Week 4: shift from cat 2 to cat 1 | 5 | 7 | 2 | 4 | 7
  Week 4: shift from cat 2 to cat 2: number analyzed (Participants) | 42 | 26 | 16 | 44 | 46
  Week 4: shift from cat 2 to cat 2 | 1 | 0 | 0 | 0 | 0
  Week 4: shift from cat 2 to cat 3: number analyzed (Participants) | 42 | 26 | 16 | 44 | 46
  Week 4: shift from cat 2 to cat 3 | 0 | 0 | 0 | 0 | 0
  Week 4: shift from cat 3 to cat 1: number analyzed (Participants) | 42 | 26 | 16 | 44 | 46
  Week 4: shift from cat 3 to cat 1 | 1 | 5 | 1 | 2 | 1
  Week 4: shift from cat 3 to cat 2: number analyzed (Participants) | 42 | 26 | 16 | 44 | 46
  Week 4: shift from cat 3 to cat 2 | 0 | 0 | 0 | 0 | 0
  Week 4: shift from cat 3 to cat 3: number analyzed (Participants) | 42 | 26 | 16 | 44 | 46
  Week 4: shift from cat 3 to cat 3 | 0 | 0 | 0 | 0 | 0
  Week 12: shift from cat 1 to cat 1: number analyzed (Participants) | 42 | 26 | 16 | 45 | 41
  Week 12: shift from cat 1 to cat 1 | 34 | 14 | 12 | 40 | 33
  Week 12: shift from cat 1 to cat 2: number analyzed (Participants) | 42 | 26 | 16 | 45 | 41
  Week 12: shift from cat 1 to cat 2 | 0 | 0 | 0 | 0 | 0
  Week 12: shift from cat 1 to cat 3: number analyzed (Participants) | 42 | 26 | 16 | 45 | 41
  Week 12: shift from cat 1 to cat 3 | 0 | 0 | 0 | 0 | 0
  Week 12: shift from cat 2 to cat 1: number analyzed (Participants) | 42 | 26 | 16 | 45 | 41
  Week 12: shift from cat 2 to cat 1 | 7 | 5 | 3 | 2 | 7
  Week 12: shift from cat 2 to cat 2: number analyzed (Participants) | 42 | 26 | 16 | 45 | 41
  Week 12: shift from cat 2 to cat 2 | 0 | 2 | 0 | 1 | 0
  Week 12: shift from cat 2 to cat 3: number analyzed (Participants) | 42 | 26 | 16 | 45 | 41
  Week 12: shift from cat 2 to cat 3 | 0 | 0 | 0 | 0 | 0
  Week 12: shift from cat 3 to cat 1: number analyzed (Participants) | 42 | 26 | 16 | 45 | 41
  Week 12: shift from cat 3 to cat 1 | 1 | 5 | 1 | 2 | 1
  Week 12: shift from cat 3 to cat 2: number analyzed (Participants) | 42 | 26 | 16 | 45 | 41
  Week 12: shift from cat 3 to cat 2 | 0 | 0 | 0 | 0 | 0
  Week 12: shift from cat 3 to cat 3: number analyzed (Participants) | 42 | 26 | 16 | 45 | 41
  Week 12: shift from cat 3 to cat 3 | 0 | 0 | 0 | 0 | 0
  Week 16: shift from cat 1 to cat 1: number analyzed (Participants) | 41 | 27 | 16 | 46 | 41
  Week 16: shift from cat 1 to cat 1 | 33 | 15 | 12 | 40 | 33
  Week 16: shift from cat 1 to cat 2: number analyzed (Participants) | 41 | 27 | 16 | 46 | 41
  Week 16: shift from cat 1 to cat 2 | 0 | 0 | 0 | 0 | 0
  Week 16: shift from cat 1 to cat 3: number analyzed (Participants) | 41 | 27 | 16 | 46 | 41
  Week 16: shift from cat 1 to cat 3 | 0 | 0 | 0 | 0 | 0
  Week 16: shift from cat 2 to cat 1: number analyzed (Participants) | 41 | 27 | 16 | 46 | 41
  Week 16: shift from cat 2 to cat 1 | 6 | 6 | 3 | 4 | 7
  Week 16: shift from cat 2 to cat 2: number analyzed (Participants) | 41 | 27 | 16 | 46 | 41
  Week 16: shift from cat 2 to cat 2 | 1 | 1 | 0 | 0 | 0
  Week 16: shift from cat 2 to cat 3: number analyzed (Participants) | 41 | 27 | 16 | 46 | 41
  Week 16: shift from cat 2 to cat 3 | 0 | 0 | 0 | 0 | 0
  Week 16: shift from cat 3 to cat 1: number analyzed (Participants) | 41 | 27 | 16 | 46 | 41
  Week 16: shift from cat 3 to cat 1 | 1 | 5 | 1 | 2 | 1
  Week 16: shift from cat 3 to cat 2: number analyzed (Participants) | 41 | 27 | 16 | 46 | 41
  Week 16: shift from cat 3 to cat 2 | 0 | 0 | 0 | 0 | 0
  Week 16: shift from cat 3 to cat 3: number analyzed (Participants) | 41 | 27 | 16 | 46 | 41
  Week 16: shift from cat 3 to cat 3 | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 for Clinical Laboratory Parameters Hematology: Erythrocytes
Description: Blood samples for clinical hematology assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: 10^12*cells/L
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
10^12*cells/L
  Baseline | 4.568 (0.392) | 4.537 (0.375) | 4.510 (0.365) | 4.516 (0.429) | 4.563 (0.406)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -0.106 (0.262) | -0.108 (0.218) | 0.007 (0.254) | -0.095 (0.215) | -0.090 (0.210)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline | -0.094 (0.278) | -0.083 (0.217) | 0.072 (0.200) | -0.087 (0.203) | -0.077 (0.229)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline | -0.057 (0.277) | -0.085 (0.256) | 0.039 (0.273) | -0.057 (0.265) | -0.057 (0.202)
  Week 16: Change from baseline: number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | -0.060 (0.293) | -0.023 (0.250) | -0.033 (0.290) | -0.085 (0.254) | -0.040 (0.240)

41. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 for Clinical Laboratory Parameters Hematology: Hematocrit
Description: Blood samples for clinical hematology assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: Volume proportion
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Volume proportion
  Baseline | 0.4230 (0.0347) | 0.4184 (0.0303) | 0.4102 (0.0384) | 0.4088 (0.0312) | 0.4182 (0.0346)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -0.0121 (0.0261) | -0.0079 (0.0220) | 0.0016 (0.0211) | -0.0079 (0.0195) | -0.0138 (0.0199)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline | -0.0097 (0.0249) | -0.0060 (0.0194) | 0.0075 (0.0144) | -0.0080 (0.0186) | -0.0100 (0.0234)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline | -0.0106 (0.0294) | -0.0036 (0.0220) | 0.0087 (0.0276) | -0.0083 (0.0258) | -0.0115 (0.0231)
  Week 16: Change from baseline: number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | -0.0140 (0.0258) | -0.0006 (0.0250) | 0.0015 (0.0244) | -0.0100 (0.0235) | -0.0099 (0.0274)

42. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 in Clinical Laboratory Parameters Hematology: Hemoglobin
Description: Blood samples for clinical hematology assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
g/L
  Baseline | 138.4 (10.9) | 137.3 (10.0) | 136.4 (11.6) | 134.6 (9.8) | 135.6 (11.4)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -3.0 (7.8) | -3.0 (6.6) | -0.2 (7.5) | -2.8 (6.3) | -2.5 (5.4)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline | -2.7 (8.1) | -2.6 (6.7) | 2.6 (5.3) | -2.8 (5.7) | -2.4 (6.2)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline | -2.1 (7.7) | -2.5 (7.5) | 0.8 (7.5) | -2.3 (7.1) | -1.5 (5.9)
  Week 16: Change from baseline: number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | -1.9 (8.5) | -0.7 (6.9) | -1.7 (8.2) | -2.6 (6.9) | -1.1 (6.4)

43. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 in Clinical Laboratory Parameters Hematology: Erythrocytes Mean Corpuscular Volume
Description: Blood samples for clinical hematology assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
fL
  Baseline | 92.74 (4.65) | 92.39 (4.51) | 90.92 (3.00) | 90.82 (5.25) | 91.88 (5.69)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -0.56 (2.35) | 0.51 (2.58) | 0.24 (2.02) | 0.10 (1.72) | -1.29 (3.35)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline | -0.22 (2.53) | 0.49 (2.31) | 0.27 (2.85) | -0.10 (1.92) | -0.73 (4.48)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline | -1.22 (3.30) | 0.98 (3.41) | 1.18 (2.72) | -0.77 (2.66) | -1.47 (4.49)
  Week 16: Change from baseline: number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline | -1.91 (2.99) | 0.36 (3.41) | 1.05 (2.39) | -0.55 (4.13) | -1.42 (5.06)

44. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 in Clinical Laboratory Parameters Hematology: Leukocytes, Platelets, Basophils, Eosinophils, Lymphocytes, Monocytes and Neutrophils
Description: Blood samples for clinical hematology assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: 10^9*cells/L
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
10^9*cells/L
  Baseline (Leukocytes) | 6.09 (1.80) | 6.17 (1.89) | 6.32 (1.35) | 6.31 (1.74) | 6.40 (1.76)
  Week 2: Change from baseline (Leukocytes): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Leukocytes) | -0.19 (1.02) | -0.24 (0.99) | -0.13 (0.97) | -0.25 (1.33) | -0.12 (1.44)
  Week 4: Change from baseline (Leukocytes): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Leukocytes) | 0.41 (2.80) | -0.09 (0.96) | 0.16 (1.02) | -0.27 (1.44) | -0.20 (1.04)
  Week 12: Change from baseline (Leukocytes): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Leukocytes) | -0.12 (1.28) | -0.11 (1.07) | 0.08 (1.98) | -0.29 (1.55) | -0.08 (1.59)
  Week 16: Change from baseline (Leukocytes): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Leukocytes) | -0.20 (1.15) | 0.19 (1.84) | -0.05 (1.20) | -0.12 (1.88) | 0.09 (1.18)
  Baseline (Platelets): number analyzed (Participants) | 47 | 31 | 17 | 51 | 52
  Baseline (Platelets) | 273.6 (53.7) | 270.8 (66.2) | 254.9 (37.2) | 280.6 (62.8) | 277.0 (59.3)
  Week 2: Change from baseline (Platelets): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Platelets) | 0.6 (36.2) | -3.9 (31.8) | -6.0 (22.4) | -5.5 (32.4) | -3.0 (30.7)
  Week 4: Change from baseline (Platelets): number analyzed (Participants) | 45 | 30 | 17 | 50 | 47
  Week 4: Change from baseline (Platelets) | 9.5 (43.7) | -2.1 (27.6) | 7.6 (35.8) | -5.7 (29.9) | -1.4 (34.4)
  Week 12: Change from baseline (Platelets): number analyzed (Participants) | 44 | 30 | 16 | 48 | 44
  Week 12: Change from baseline (Platelets) | 8.2 (54.7) | -0.5 (33.1) | 14.7 (23.9) | 0.0 (30.6) | 1.3 (45.7)
  Week16: Change from baseline (Platelets): number analyzed (Participants) | 41 | 30 | 16 | 50 | 45
  Week16: Change from baseline (Platelets) | 12.4 (28.6) | 5.7 (37.3) | 3.9 (28.7) | 1.2 (32.9) | 9.5 (38.0)
  Baseline (Basophils) | 0.03 (0.04) | 0.05 (0.05) | 0.04 (0.05) | 0.03 (0.05) | 0.03 (0.04)
  Week 2: Change from baseline (Basophils): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Basophils) | 0.00 (0.04) | 0.00 (0.02) | -0.02 (0.04) | 0.00 (0.04) | 0.01 (0.04)
  Week 4: Change from baseline (Basophils): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Basophils) | 0.00 (0.05) | -0.01 (0.03) | -0.02 (0.04) | -0.01 (0.04) | 0.01 (0.05)
  Week 12: Change from baseline (Basophils): number analyzed (Participants) | 44 | 30 | 15 | 49 | 44
  Week 12: Change from baseline (Basophils) | 0.00 (0.04) | -0.01 (0.04) | -0.02 (0.06) | 0.00 (0.05) | 0.00 (0.03)
  Week 16: Change from baseline (Basophils): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Basophils) | 0.00 (0.04) | 0.00 (0.00) | 0.00 (0.05) | -0.01 (0.04) | 0.01 (0.05)
  Baseline (Eosinophils) | 0.14 (0.09) | 0.19 (0.12) | 0.18 (0.15) | 0.20 (0.24) | 0.18 (0.14)
  Week 2: Change from baseline (Eosinophils): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Eosinophils) | 0.00 (0.06) | 0.00 (0.09) | -0.01 (0.07) | -0.03 (0.12) | -0.02 (0.09)
  Week 4: Change from baseline (Eosinophils): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Eosinophils) | -0.01 (0.09) | -0.01 (0.08) | -0.01 (0.11) | -0.03 (0.16) | -0.02 (0.07)
  Week 12: Change from baseline (Eosinophils): number analyzed (Participants) | 44 | 30 | 15 | 49 | 44
  Week 12: Change from baseline (Eosinophils) | 0.02 (0.09) | 0.02 (0.09) | 0.00 (0.11) | -0.05 (0.19) | -0.03 (0.09)
  Week 16: Change from baseline (Eosinophils): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Eosinophils) | 0.00 (0.10) | -0.02 (0.08) | -0.01 (0.13) | -0.05 (0.17) | -0.02 (0.11)
  Baseline (Lymphocytes) | 1.98 (0.67) | 1.90 (0.63) | 1.78 (0.50) | 2.11 (0.66) | 2.00 (0.62)
  Week 2: Change from baseline (Lymphocytes): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Lymphocytes) | -0.06 (0.34) | -0.11 (0.33) | -0.10 (0.31) | -0.11 (0.41) | -0.14 (0.39)
  Week 4: Change from baseline (Lymphocytes): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Lymphocytes) | -0.08 (0.38) | -0.13 (0.34) | 0.04 (0.45) | -0.08 (0.50) | -0.02 (0.38)
  Week 12: Change from baseline (Lymphocytes): number analyzed (Participants) | 44 | 30 | 15 | 49 | 44
  Week 12: Change from baseline (Lymphocytes) | -0.05 (0.36) | -0.08 (0.34) | -0.07 (0.24) | -0.09 (0.47) | -0.05 (0.29)
  Week 16: Change from baseline (Lymphocytes): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Lymphocytes) | -0.14 (0.46) | -0.11 (0.40) | -0.07 (0.32) | -0.13 (0.39) | 0.01 (0.36)
  Baseline (Monocytes) | 0.44 (0.13) | 0.47 (0.14) | 0.51 (0.10) | 0.47 (0.14) | 0.46 (0.17)
  Week 2: Change from baseline (Monocytes): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Monocytes) | 0.00 (0.09) | -0.02 (0.13) | -0.02 (0.13) | -0.05 (0.14) | -0.01 (0.11)
  Week 4: Change from baseline (Monocytes): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Monocytes) | 0.02 (0.09) | -0.03 (0.10) | 0.01 (0.12) | -0.03 (0.11) | -0.02 (0.12)
  Week 12: Change from baseline (Monocytes): number analyzed (Participants) | 44 | 30 | 15 | 49 | 44
  Week 12: Change from baseline (Monocytes) | 0.01 (0.11) | -0.03 (0.10) | -0.06 (0.11) | -0.03 (0.13) | 0.00 (0.15)
  Week 16: Change from baseline (Monocytes): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Monocytes) | 0.01 (0.11) | -0.02 (0.14) | -0.03 (0.13) | 0.00 (0.13) | 0.00 (0.14)
  Baseline (Neutrophils) | 3.50 (1.34) | 3.59 (1.33) | 3.81 (1.13) | 3.51 (1.41) | 3.73 (1.28)
  Week 2: Change from baseline (Neutrophils): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Neutrophils) | -0.14 (0.79) | -0.15 (0.84) | 0.03 (0.80) | -0.08 (1.24) | 0.01 (1.32)
  Week 4: Change from baseline (Neutrophils): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Neutrophils) | 0.11 (1.04) | 0.09 (0.86) | 0.14 (0.70) | -0.13 (1.24) | -0.16 (0.91)
  Week 12: Change from baseline (Neutrophils): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Neutrophils) | -0.11 (1.16) | -0.02 (0.97) | 0.22 (1.79) | -0.13 (1.26) | -0.01 (1.39)
  Week 16: Change from baseline (Neutrophils): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Neutrophils) | -0.08 (1.19) | 0.33 (1.70) | 0.05 (0.96) | 0.04 (1.73) | 0.10 (0.95)

45. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 in Clinical Laboratory Parameters Hematology: Leukocytes, Basophils, Eosinophils, Lymphocytes, Monocytes and Neutrophils
Description: Blood samples for clinical hematology assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: Percentage of total white blood cells
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Percentage of total white blood cells
  Baseline (Basophils/ Leukocytes) | 0.61 (0.36) | 0.72 (0.34) | 0.59 (0.26) | 0.69 (0.47) | 0.59 (0.31)
  Week 2: Change from baseline (Basophils/ Leukocytes): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Basophils/ Leukocytes) | 0.02 (0.22) | -0.01 (0.19) | -0.01 (0.18) | -0.04 (0.30) | 0.07 (0.20)
  Week 4: Change from baseline (Basophils/ Leukocytes): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Basophils/ Leukocytes) | 0.03 (0.28) | -0.04 (0.21) | -0.02 (0.22) | -0.06 (0.31) | 0.08 (0.30)
  Week 12: Change from baseline (Basophils/ Leukocytes): number analyzed (Participants) | 44 | 30 | 15 | 49 | 44
  Week 12: Change from baseline (Basophils/ Leukocytes) | 0.02 (0.35) | 0.01 (0.26) | 0.03 (0.15) | -0.07 (0.31) | 0.05 (0.21)
  Week 16: Change from baseline (Basophils/ Leukocytes): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Basophils/ Leukocytes) | 0.00 (0.27) | 0.05 (0.20) | 0.06 (0.22) | -0.05 (0.32) | 0.01 (0.19)
  Baseline (Eosinophils/ Leukocytes) | 2.17 (1.22) | 2.89 (1.67) | 2.66 (1.80) | 2.97 (3.43) | 2.76 (1.78)
  Week 2: Change from baseline (Eosinophils/ Leukocytes): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Eosinophils/ Leukocytes) | 0.16 (0.87) | 0.20 (1.01) | -0.12 (0.75) | -0.24 (1.78) | -0.13 (1.17)
  Week 4: Change from baseline (Eosinophils/ Leukocytes): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Eosinophils/ Leukocytes) | -0.13 (0.84) | -0.06 (0.99) | -0.15 (1.14) | -0.43 (2.43) | -0.17 (0.99)
  Week 12: Change from baseline (Eosinophils/ Leukocytes): number analyzed (Participants) | 44 | 30 | 15 | 49 | 44
  Week 12: Change from baseline (Eosinophils/ Leukocytes) | 0.33 (1.22) | 0.41 (1.49) | 0.11 (1.16) | -0.53 (2.58) | -0.27 (1.43)
  Week16: Change from baseline (Eosinophils/ Leukocytes): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week16: Change from baseline (Eosinophils/ Leukocytes) | 0.10 (1.59) | -0.15 (1.18) | 0.00 (1.53) | -0.42 (2.33) | -0.32 (1.57)
  Baseline (Lymphocytes/ Leukocytes) | 32.87 (7.02) | 31.31 (6.31) | 28.71 (7.07) | 34.20 (9.42) | 31.95 (7.49)
  Week 2: Change from baseline (Lymphocytes/ Leukocytes): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Lymphocytes/ Leukocytes) | 0.27 (5.12) | -0.54 (5.60) | -1.32 (4.45) | -0.83 (7.48) | -1.37 (6.02)
  Week 4: Change from baseline (Lymphocytes/ Leukocytes): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Lymphocytes/ Leukocytes) | -1.24 (5.98) | -1.25 (5.12) | -0.89 (3.68) | -0.43 (7.03) | 0.68 (4.85)
  Week 12: Change from baseline (Lymphocytes/ Leukocytes): number analyzed (Participants) | 44 | 30 | 15 | 49 | 44
  Week 12: Change from baseline (Lymphocytes/ Leukocytes) | -0.32 (6.82) | -0.51 (6.59) | 0.13 (4.78) | -0.41 (6.56) | -0.07 (4.94)
  Week 16: Change from baseline (Lymphocytes/ Leukocytes): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Lymphocytes/ Leukocytes) | -0.89 (7.90) | -1.40 (8.07) | -0.75 (4.70) | -0.95 (7.10) | -0.70 (4.39)
  Baseline (Monocytes/Leukocytes) | 7.41 (1.76) | 7.71 (2.07) | 8.18 (1.62) | 7.55 (1.67) | 7.15 (1.67)
  Week 2: Change from baseline (Monocytes/Leukocytes): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Monocytes/Leukocytes) | 0.19 (1.11) | 0.05 (1.83) | -0.24 (2.01) | -0.36 (1.59) | 0.08 (1.20)
  Week 4: Change from baseline (Monocytes/Leukocytes): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Monocytes/Leukocytes) | 0.24 (1.31) | -0.19 (1.24) | -0.29 (1.71) | -0.13 (1.25) | 0.21 (1.81)
  Week 12: Change from baseline (Monocytes/Leukocytes): number analyzed (Participants) | 44 | 30 | 15 | 49 | 44
  Week 12: Change from baseline (Monocytes/Leukocytes) | 0.45 (1.34) | -0.19 (1.64) | -0.67 (1.27) | -0.01 (1.57) | 0.24 (1.52)
  Week 16: Change from baseline (Monocytes/Leukocytes): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Monocytes/Leukocytes) | 0.48 (1.67) | -0.50 (1.75) | -0.48 (1.45) | 0.27 (1.67) | 0.08 (1.68)
  Baseline (Neutrophils/Leukocytes) | 56.93 (8.12) | 57.37 (7.13) | 59.85 (8.07) | 54.59 (0.43) | 57.56 (8.01)
  Week 2: Change from baseline (Neutrophils/Leukocytes): number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline (Neutrophils/Leukocytes) | -0.64 (6.11) | 0.29 (6.64) | 1.70 (5.11) | 1.47 (8.32) | 1.36 (6.75)
  Week 4: Change from baseline (Neutrophils/Leukocytes): number analyzed (Participants) | 45 | 30 | 17 | 51 | 47
  Week 4: Change from baseline (Neutrophils/Leukocytes) | 1.10 (6.92) | 1.54 (5.78) | 1.35 (4.76) | 1.05 (8.38) | -0.80 (6.01)
  Week 12: Change from baseline (Neutrophils/Leukocytes): number analyzed (Participants) | 44 | 30 | 15 | 49 | 44
  Week 12: Change from baseline (Neutrophils/Leukocytes) | -0.48 (7.92) | 0.27 (7.61) | 0.40 (5.40) | 1.01 (7.54) | 0.05 (5.60)
  Week 16: Change from baseline (Neutrophils/Leukocytes): number analyzed (Participants) | 41 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Neutrophils/Leukocytes) | 0.30 (9.57) | 2.00 (9.27) | 1.17 (5.31) | 1.14 (8.14) | 0.94 (5.30)

46. Secondary Outcome: Change From Baseline at Weeks 2, 4, 8, 12 and 16 in Clinical Laboratory Parameters Biochemistry: Sodium, Potassium, Glucose, Urea Nitrogen, Calcium, Phosphate, Bicarbonate, Magnesium and Chloride
Description: Blood samples for clinical chemistry assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
mmol/L
  Baseline (Sodium) | 141.3 (2.0) | 141.6 (2.4) | 141.6 (2.9) | 141.2 (1.8) | 141.3 (2.0)
  Week 2: Change from baseline (Sodium): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Sodium) | -0.1 (1.9) | 0.1 (2.1) | -0.6 (2.0) | -0.5 (1.8) | -0.5 (1.7)
  Week 4: Change from baseline (Sodium): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Sodium) | -0.5 (1.7) | -0.2 (2.1) | -0.9 (2.4) | -0.3 (1.8) | 0.0 (1.6)
  Week 8: Change from baseline (Sodium): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Sodium) | 0.0 (1.8) | -0.8 (2.5) | -0.6 (1.6) | 0.1 (2.0) | 0.1 (1.7)
  Week 12: Change from baseline (Sodium): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Sodium) | -0.5 (1.9) | -0.6 (2.5) | -0.9 (1.7) | 0.0 (2.2) | -0.1 (1.8)
  Week 16: Change from baseline (Sodium): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Sodium) | -0.2 (1.7) | -0.1 (2.1) | -0.1 (2.0) | -0.2 (2.0) | -0.3 (1.8)
  Baseline (Potassium) | 4.51 (0.38) | 4.43 (0.30) | 4.23 (0.33) | 4.37 (0.44) | 4.36 (0.45)
  Week 2: Change from baseline (Potassium): number analyzed (Participants) | 43 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Potassium) | -0.02 (0.35) | -0.08 (0.36) | 0.06 (0.35) | 0.01 (0.44) | -0.07 (0.40)
  Week 4: Change from baseline (Potassium): number analyzed (Participants) | 45 | 31 | 17 | 50 | 47
  Week 4: Change from baseline (Potassium) | -0.04 (0.39) | -0.09 (0.40) | 0.06 (0.27) | -0.02 (0.45) | -0.13 (0.31)
  Week 8: Change from baseline (Potassium): number analyzed (Participants) | 41 | 30 | 13 | 50 | 43
  Week 8: Change from baseline (Potassium) | 0.06 (0.39) | -0.10 (0.34) | -0.05 (0.30) | 0.02 (0.51) | -0.11 (0.42)
  Week 12: Change from baseline (Potassium): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Potassium) | -0.10 (0.40) | -0.07 (0.34) | 0.10 (0.41) | 0.03 (0.51) | -0.16 (0.40)
  Week 16: Change from baseline (Potassium): number analyzed (Participants) | 43 | 30 | 16 | 51 | 44
  Week 16: Change from baseline (Potassium) | -0.13 (0.39) | -0.10 (0.33) | -0.04 (0.33) | 0.04 (0.45) | -0.16 (0.40)
  Baseline (Glucose) | 5.06 (0.83) | 5.32 (1.11) | 5.16 (0.71) | 5.04 (0.74) | 5.81 (2.70)
  Week 2: Change from baseline (Glucose): number analyzed (Participants) | 43 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Glucose) | 0.22 (1.12) | -0.07 (0.92) | 0.04 (1.01) | 0.28 (0.97) | 0.21 (1.89)
  Week 4: Change from baseline (Glucose): number analyzed (Participants) | 45 | 31 | 17 | 51 | 47
  Week 4: Change from baseline (Glucose) | 0.24 (0.73) | 0.02 (0.87) | -0.24 (1.08) | 0.02 (0.87) | -0.29 (2.39)
  Week 8: Change from baseline (Glucose): number analyzed (Participants) | 41 | 30 | 13 | 50 | 43
  Week 8: Change from baseline (Glucose) | 0.12 (0.54) | -0.15 (1.15) | -0.13 (1.17) | 0.01 (1.09) | -0.12 (1.35)
  Week 12: Change from baseline (Glucose): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Glucose) | -0.06 (0.94) | -0.09 (1.06) | 0.13 (0.55) | 0.21 (1.48) | -0.34 (1.82)
  Week 16: Change from baseline (Glucose): number analyzed (Participants) | 43 | 30 | 16 | 51 | 44
  Week 16: Change from baseline (Glucose) | 0.14 (0.81) | 0.06 (1.03) | 0.10 (0.94) | 0.09 (1.02) | -0.43 (1.58)
  Baseline (Urea Nitrogen) | 5.74 (1.49) | 5.64 (1.54) | 5.70 (1.45) | 5.34 (1.51) | 5.31 (1.26)
  Week 2: Change from baseline (Urea Nitrogen): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Urea Nitrogen) | -0.43 (1.05) | 0.04 (1.21) | 0.50 (1.35) | 0.50 (1.25) | 0.24 (1.15)
  Week 4: Change from baseline (Urea Nitrogen): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Urea Nitrogen) | -0.30 (1.58) | 0.12 (0.95) | 0.17 (1.25) | 0.36 (1.42) | 0.12 (1.22)
  Week 8: Change from baseline (Urea Nitrogen): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Urea Nitrogen) | -0.23 (1.10) | -0.34 (1.18) | 0.13 (1.71) | 0.53 (1.58) | -0.03 (1.34)
  Week 12: Change from baseline (Urea Nitrogen): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Urea Nitrogen) | -0.21 (1.20) | -0.17 (1.13) | 0.45 (2.11) | 0.31 (1.09) | -0.10 (1.31)
  Week 16: Change from baseline (Urea Nitrogen): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Urea Nitrogen) | -0.24 (1.41) | -0.19 (1.32) | -0.03 (1.57) | 0.24 (1.11) | -0.01 (1.25)
  Baseline (Calcium) | 2.348 (0.082) | 2.354 (0.093) | 2.325 (0.091) | 2.347 (0.117) | 2.342 (0.091)
  Week 2: Change from baseline (Calcium): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Calcium) | -0.046 (0.081) | -0.052 (0.082) | 0.011 (0.102) | -0.019 (0.079) | -0.050 (0.101)
  Week 4: Change from baseline (Calcium): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Calcium) | -0.035 (0.094) | -0.035 (0.077) | 0.028 (0.068) | -0.018 (0.099) | -0.036 (0.094)
  Week 8: Change from baseline (Calcium): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Calcium) | -0.008 (0.109) | -0.034 (0.085) | 0.002 (0.091) | -0.021 (0.108) | -0.042 (0.077)
  Week 12: Change from baseline (Calcium): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Calcium) | -0.006 (0.088) | -0.018 (0.091) | 0.014 (0.108) | -0.014 (0.097) | -0.042 (0.084)
  Week 16 Change from baseline (Calcium): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16 Change from baseline (Calcium) | -0.005 (0.090) | -0.033 (0.093) | 0.003 (0.097) | -0.009 (0.100) | -0.027 (0.104)
  Baseline (Phosphate) | 1.28 (0.15) | 1.28 (0.15) | 1.17 (0.15) | 1.26 (0.16) | 1.22 (0.15)
  Week 2: Change from baseline (Phosphate): number analyzed (Participants) | 43 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Phosphate) | -0.02 (0.13) | 0.00 (0.13) | 0.03 (0.15) | 0.00 (0.15) | -0.02 (0.17)
  Week 4: Change from baseline (Phosphate): number analyzed (Participants) | 45 | 31 | 17 | 50 | 47
  Week 4: Change from baseline (Phosphate) | 0.00 (0.14) | 0.00 (0.16) | 0.05 (0.09) | -0.01 (0.15) | -0.03 (0.15)
  Week 8: Change from baseline (Phosphate) | -0.01 (0.13) | -0.02 (0.15) | 0.07 (0.11) | 0.02 (0.18) | -0.02 (0.14)
  Week 12: Change from baseline (Phosphate): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Phosphate) | -0.02 (0.16) | -0.02 (0.17) | 0.06 (0.15) | 0.02 (0.19) | -0.06 (0.14)
  Week 16: Change from baseline (Phosphate): number analyzed (Participants) | 43 | 30 | 16 | 51 | 44
  Week 16: Change from baseline (Phosphate) | -0.02 (0.17) | -0.01 (0.16) | 0.00 (0.14) | -0.01 (0.17) | -0.01 (0.13)
  Baseline (Bicarbonate) | 25.5 (2.4) | 26.6 (3.4) | 26.2 (3.7) | 26.7 (2.7) | 26.0 (2.9)
  Week 2: Change from baseline (Bicarbonate): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Bicarbonate) | 0.3 (1.7) | 0.0 (2.0) | -0.6 (2.3) | -0.5 (2.1) | -0.2 (2.0)
  Week 4: Change from baseline (Bicarbonate): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Bicarbonate) | 0.2 (2.0) | -0.1 (2.0) | -0.1 (2.3) | -0.4 (2.1) | 0.0 (1.7)
  Week 8: Change from baseline (Bicarbonate): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Bicarbonate) | 0.3 (1.8) | 0.0 (2.3) | -0.2 (2.1) | -0.6 (1.9) | 0.3 (1.9)
  Week 12: Change from baseline (Bicarbonate): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Bicarbonate) | 0.6 (2.1) | -0.4 (2.1) | -0.5 (2.4) | -0.6 (1.9) | -0.2 (1.9)
  Week 16: Change from baseline (Bicarbonate): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Bicarbonate) | 0.4 (1.5) | -0.1 (2.3) | -0.5 (2.7) | -0.3 (2.3) | -0.1 (2.1)
  Baseline (Magnesium) | 0.809 (0.075) | 0.833 (0.084) | 0.826 (0.075) | 0.821 (0.067) | 0.817 (0.076)
  Week 2: Change from baseline (Magnesium): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Magnesium) | -0.011 (0.066) | -0.027 (0.070) | -0.009 (0.065) | -0.013 (0.066) | -0.037 (0.057)
  Week 4: Change from baseline (Magnesium): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Magnesium) | -0.008 (0.054) | -0.035 (0.057) | 0.002 (0.052) | -0.017 (0.061) | -0.017 (0.060)
  Week 8: Change from baseline (Magnesium): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Magnesium) | 0.005 (0.056) | -0.016 (0.065) | 0.010 (0.048) | 0.005 (0.077) | -0.008 (0.063)
  Week 12: Change from baseline (Magnesium): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Magnesium) | -0.033 (0.059) | -0.025 (0.060) | -0.035 (0.058) | -0.012 (0.070) | -0.016 (0.059)
  Week 16: Change from baseline (Magnesium): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Magnesium) | -0.024 (0.052) | -0.043 (0.069) | -0.022 (0.063) | -0.025 (0.057) | -0.022 (0.052)
  Baseline (Chloride) | 105.6 (2.2) | 105.4 (2.1) | 105.5 (2.4) | 104.8 (2.4) | 105.3 (2.6)
  Week 2: Change from baseline (Chloride): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Chloride) | 0.2 (2.0) | 0.3 (2.2) | 0.3 (2.2) | 0.5 (2.2) | -0.1 (1.9)
  Week 4: Change from baseline (Chloride): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Chloride) | -0.3 (1.7) | -0.2 (1.8) | -0.7 (2.5) | 0.3 (2.2) | 0.2 (2.1)
  Week 8: Change from baseline (Chloride): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Chloride) | 0.2 (1.9) | -0.3 (2.0) | -0.4 (1.8) | 0.5 (2.3) | 0.3 (1.6)
  Week 12: Change from baseline (Chloride): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Chloride) | -0.5 (2.2) | -0.1 (2.2) | -0.3 (1.9) | 0.5 (2.3) | 0.8 (2.0)
  Week 16: Change from baseline (Chloride): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Chloride) | -0.5 (1.8) | 0.2 (2.2) | 0.6 (2.6) | 0.1 (1.9) | 0.1 (2.2)

47. Secondary Outcome: Change From Baseline at Weeks 2, 4, 8, 12 and 16 in Clinical Laboratory Parameters Biochemistry: Creatinine and Bilirubin
Description: Blood samples for clinical chemistry assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
umol/L
  Baseline (Creatinine) | 68.8 (11.2) | 68.5 (11.7) | 68.1 (14.9) | 71.4 (11.3) | 70.1 (11.9)
  Week 2: Change from baseline (Creatinine): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Creatinine) | 0.8 (7.2) | -0.2 (8.9) | 2.9 (9.7) | 0.7 (6.5) | 0.6 (7.0)
  Week 4: Change from baseline (Creatinine): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Creatinine) | -0.9 (6.0) | 0.6 (8.1) | 2.7 (9.8) | 1.9 (7.8) | 0.2 (7.8)
  Week 8: Change from baseline (Creatinine): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Creatinine) | 1.0 (6.3) | -1.0 (7.8) | 4.8 (5.3) | 0.6 (7.8) | 0.5 (9.0)
  Week 12: Change from baseline (Creatinine): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Creatinine) | 0.7 (8.9) | 2.1 (7.7) | 4.2 (11.2) | -0.5 (7.4) | -2.8 (8.0)
  Week 16: Change from baseline (Creatinine): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Creatinine) | 0.1 (7.6) | 1.5 (6.9) | 6.5 (8.5) | -0.9 (8.2) | -0.2 (12.9)
  Baseline (Bilirubin) | 9.1 (4.1) | 8.4 (2.9) | 8.9 (3.1) | 9.6 (5.0) | 8.1 (2.8)
  Week 2: Change from baseline (Bilirubin): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Bilirubin) | -0.5 (2.2) | 0.1 (2.2) | 1.4 (2.0) | 1.1 (3.3) | 1.7 (2.5)
  Week 4: Change from baseline (Bilirubin): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Bilirubin) | -0.2 (2.6) | 0.4 (2.7) | 2.3 (2.8) | 1.0 (3.3) | 1.3 (3.0)
  Week 8: Change from baseline (Bilirubin): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Bilirubin) | -0.1 (2.8) | 0.1 (2.1) | 1.8 (2.1) | 0.3 (3.1) | 0.9 (2.6)
  Week 12: Change from baseline (Bilirubin): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Bilirubin) | -0.1 (2.4) | 0.7 (2.4) | 0.8 (2.7) | -0.2 (3.8) | 1.0 (2.7)
  Week 16: Change from baseline (Bilirubin): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Bilirubin) | 0.2 (2.4) | -0.3 (3.4) | 0.8 (2.8) | -0.8 (3.7) | -0.4 (2.5)

48. Secondary Outcome: Change From Baseline at Weeks 2, 4, 8, 12 and 16 in Clinical Laboratory Parameters Biochemistry: Creatinine Kinase, Alkaline Phosphatase, Aspartate Aminotransferase, Alanine Aminotransferase and Gamma Glutamyl Transferase
Description: Blood samples for clinical chemistry assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
U/L
  Baseline (Creatine Kinase) | 102.5 (117.2) | 91.6 (55.6) | 104.2 (62.0) | 161.8 (291.4) | 139.8 (159.3)
  Week 2: Change from baseline (Creatine Kinase): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Creatine Kinase) | 28.2 (161.8) | 7.1 (45.5) | 8.7 (59.6) | -39.2 (280.5) | -44.3 (154.1)
  Week 4: Change from baseline (Creatine Kinase): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Creatine Kinase) | -1.3 (36.8) | 2.7 (23.4) | 4.3 (44.2) | -30.2 (293.1) | -40.1 (163.0)
  Week 8: Change from baseline (Creatine Kinase): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Creatine Kinase) | 15.5 (106.6) | 30.6 (127.3) | 158.1 (580.1) | -36.9 (275.8) | 4.0 (76.1)
  Week 12: Change from baseline (Creatine Kinase): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Creatine Kinase) | 7.2 (49.7) | 16.1 (44.7) | 11.7 (116.5) | -13.3 (77.4) | -40.3 (174.5)
  Week 16: Change from baseline (Creatine Kinase): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Creatine Kinase) | 7.3 (37.3) | 3.2 (34.3) | 5.6 (54.8) | -48.8 (267.0) | -44.1 (172.2)
  Baseline (Alkaline Phosphatase) | 79.8 (24.1) | 85.9 (18.4) | 80.6 (19.4) | 91.3 (43.4) | 86.1 (25.5)
  Week 2: Change from baseline (Alkaline Phosphatase): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Alkaline Phosphatase) | -1.5 (8.4) | -1.9 (14.6) | -2.2 (6.3) | -2.5 (6.7) | -3.0 (8.2)
  Week 4: Change from baseline (Alkaline Phosphatase): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Alkaline Phosphatase) | -1.1 (6.1) | -5.2 (8.6) | 3.2 (13.1) | -3.8 (8.1) | -4.1 (8.8)
  Week 8: Change from baseline (Alkaline Phosphatase): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Alkaline Phosphatase) | -2.0 (8.5) | -5.0 (10.8) | -1.0 (6.2) | -5.1 (10.8) | -4.5 (12.0)
  Week 12: Change from baseline (Alkaline Phosphatase): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Alkaline Phosphatase) | -0.5 (8.2) | -3.2 (8.9) | 0.2 (11.5) | -4.4 (11.8) | -4.5 (8.1)
  Week 16: Change from baseline (Alkaline Phosphatase): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Alkaline Phosphatase) | -0.1 (8.5) | -0.6 (14.2) | -4.9 (10.4) | -0.1 (9.6) | -2.6 (8.0)
  Baseline (Aspartate Aminotransferase) | 24.7 (6.0) | 24.4 (6.5) | 24.4 (5.1) | 24.8 (8.0) | 24.9 (6.0)
  Week 2: Change from baseline (Aspartate Aminotransferase): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Aspartate Aminotransferase) | 0.9 (7.1) | 0.0 (4.0) | 0.1 (4.2) | -2.0 (7.6) | -2.3 (6.1)
  Week 4: Change from baseline (Aspartate Aminotransferase): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Aspartate Aminotransferase) | 1.5 (6.3) | -0.2 (3.8) | 4.6 (17.7) | -1.8 (6.7) | -0.3 (6.9)
  Week 8: Change from baseline (Aspartate Aminotransferase): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Aspartate Aminotransferase) | -1.3 (5.0) | -0.5 (4.7) | 3.4 (24.2) | -1.8 (6.9) | -1.2 (5.2)
  Week 12: Change from baseline (Aspartate Aminotransferase): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Aspartate Aminotransferase) | -1.1 (4.3) | 0.3 (3.5) | 0.9 (8.1) | -1.8 (4.7) | -2.0 (7.6)
  Week 16: Change from baseline (Aspartate Aminotransferase): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Aspartate Aminotransferase) | 0.7 (5.1) | 0.9 (7.5) | -2.4 (3.6) | -0.2 (8.5) | -2.2 (5.3)
  Baseline (Alanine Aminotransferase) | 27.0 (8.7) | 24.0 (7.6) | 23.9 (10.0) | 24.4 (10.0) | 25.9 (9.0)
  Week 2: Change from baseline (Alanine Aminotransferase): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Alanine Aminotransferase) | 0.8 (10.6) | -0.1 (5.1) | -0.7 (5.6) | -2.1 (6.7) | -3.0 (7.6)
  Week 4: Change from baseline (Alanine Aminotransferase): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Alanine Aminotransferase) | 3.5 (11.6) | -1.0 (5.5) | 16.4 (70.2) | -2.1 (5.3) | -1.1 (9.5)
  Week 8: Change from baseline (Alanine Aminotransferase): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Alanine Aminotransferase) | -0.7 (6.1) | -0.3 (5.2) | 0.6 (12.2) | -0.4 (9.2) | -0.7 (10.6)
  Week 12: Change from baseline (Alanine Aminotransferase): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Alanine Aminotransferase) | -0.5 (7.4) | 0.7 (6.0) | 4.3 (21.0) | -0.6 (6.8) | -1.2 (9.1)
  Week 16: Change from baseline (Alanine Aminotransferase): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Alanine Aminotransferase) | 2.5 (13.1) | 2.0 (9.1) | -3.5 (6.9) | 3.1 (12.0) | -2.4 (6.7)
  Baseline (Gamma Glutamyl Transferase ) | 24.6 (17.4) | 25.1 (15.0) | 19.3 (15.3) | 25.5 (23.2) | 25.9 (28.0)
  Week 2: Change from baseline (Gamma Glutamyl Transferase): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Gamma Glutamyl Transferase) | -0.2 (11.3) | 0.0 (7.1) | -1.9 (6.7) | -2.7 (8.4) | -1.0 (7.6)
  Week 4: Change from baseline (Gamma Glutamyl Transferase): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Gamma Glutamyl Transferase) | 3.0 (14.8) | -0.6 (9.1) | 3.6 (14.7) | -3.5 (10.6) | 1.4 (14.6)
  Week 8: Change from baseline (Gamma Glutamyl Transferase): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Gamma Glutamyl Transferase) | -1.5 (6.4) | 0.1 (9.2) | 0.6 (5.9) | -2.8 (13.6) | 3.3 (22.6)
  Week 12: Change from baseline (Gamma Glutamyl Transferase): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Gamma Glutamyl Transferase) | -1.2 (10.7) | 1.5 (9.8) | 4.8 (13.2) | -3.0 (14.3) | 1.3 (16.2)
  Week 16: Change from baseline (Gamma Glutamyl Transferase): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Gamma Glutamyl Transferase) | -0.7 (8.8) | 2.2 (10.1) | 1.8 (14.4) | -0.7 (10.1) | -0.2 (16.4)

49. Secondary Outcome: Change From Baseline at Weeks 2, 4, 8, 12 and 16 in Clinical Laboratory Parameters Biochemistry: Protein and Albumin
Description: Blood samples for clinical chemistry assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
g/L
  Baseline (Protein) | 67.4 (4.0) | 67.5 (4.3) | 66.5 (5.1) | 67.7 (4.3) | 67.0 (4.7)
  Week 2: Change from baseline (Protein): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Protein) | -1.7 (2.9) | -2.1 (4.6) | -0.4 (3.7) | -1.5 (2.9) | -2.1 (3.7)
  Week 4: Change from baseline (Protein): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Protein) | -1.8 (3.0) | -1.5 (4.1) | 0.2 (3.3) | -1.6 (2.7) | -1.5 (3.5)
  Week 8: Change from baseline (Protein): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Protein) | -1.5 (3.4) | -2.3 (4.2) | -1.7 (4.2) | -2.0 (3.8) | -2.4 (3.3)
  Week 12: Change from baseline (Protein): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Protein) | -1.5 (3.0) | -1.5 (3.9) | -0.7 (4.6) | -1.7 (3.4) | -1.8 (3.2)
  Week 16: Change from baseline (Protein): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Protein) | -1.0 (3.2) | -1.6 (4.1) | -1.9 (5.0) | -1.8 (3.7) | -1.7 (4.0)
  Baseline (Albumin) | 44.7 (2.1) | 44.9 (2.8) | 43.6 (2.4) | 45.2 (2.4) | 44.2 (3.0)
  Week 2: Change from baseline (Albumin): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Albumin) | -1.3 (1.9) | -1.4 (2.6) | -0.1 (2.4) | -0.9 (1.8) | -1.3 (2.4)
  Week 4: Change from baseline (Albumin): number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline (Albumin) | -0.9 (2.1) | -1.0 (2.3) | 0.5 (2.2) | -0.8 (1.9) | -0.7 (2.6)
  Week 8: Change from baseline (Albumin): number analyzed (Participants) | 41 | 30 | 14 | 50 | 43
  Week 8: Change from baseline (Albumin) | -0.8 (2.2) | -1.2 (2.7) | -0.9 (2.5) | -0.8 (2.6) | -1.3 (2.2)
  Week 12: Change from baseline (Albumin): number analyzed (Participants) | 44 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Albumin) | -0.6 (1.9) | -0.7 (2.1) | 0.3 (2.6) | -0.6 (2.5) | -0.7 (2.2)
  Week 16: Change from baseline (Albumin): number analyzed (Participants) | 43 | 30 | 16 | 51 | 45
  Week 16: Change from baseline (Albumin) | 0.0 (2.0) | -0.4 (2.0) | 0.1 (3.1) | -0.6 (2.3) | -0.4 (2.8)

50. Secondary Outcome: Change From Baseline at Weeks 2, 4, 8, 12 and 16 in Clinical Laboratory Parameters Biochemistry: Hemoglobin A1C
Description: Blood samples for clinical chemistry assessment were collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 8, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
mmol/mol
  Baseline | 39.22 (8.09) | 39.05 (5.82) | 35.84 (3.39) | 38.78 (5.65) | 40.88 (10.97)
  Week 2: Change from baseline: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2: Change from baseline | -0.42 (1.46) | 0.04 (1.18) | 0.19 (1.46) | -0.08 (1.35) | -0.21 (2.32)
  Week 4: Change from baseline: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4: Change from baseline | -0.29 (1.91) | 0.00 (1.96) | 0.06 (1.47) | -0.02 (1.55) | -0.43 (4.24)
  Week 8: Change from baseline: number analyzed (Participants) | 41 | 30 | 14 | 49 | 43
  Week 8: Change from baseline | -0.40 (2.38) | 0.26 (2.16) | 0.62 (2.13) | -0.13 (1.72) | -0.28 (5.11)
  Week 12: Change from baseline: number analyzed (Participants) | 44 | 30 | 16 | 50 | 44
  Week 12: Change from baseline | 0.07 (1.96) | 0.84 (3.01) | 1.57 (2.46) | 0.55 (2.30) | -0.94 (5.33)
  Week 16: Change from baseline: number analyzed (Participants) | 43 | 30 | 16 | 51 | 44
  Week 16: Change from baseline | -0.64 (2.41) | 0.69 (2.64) | 1.16 (2.13) | -0.04 (2.22) | -1.07 (5.65)

51. Secondary Outcome: Change From Baseline at Weeks 12 and 16 in Clinical Laboratory Parameters Bone: Bone Specific Alkaline Phosphatase and Procollagen 1 N-Terminal Propeptide
Description: Blood for assessment of bone turnover markers was collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
ug/L
  Baseline (Bone Specific Alkaline Phosphatase): number analyzed (Participants) | 47 | 30 | 17 | 48 | 52
  Baseline (Bone Specific Alkaline Phosphatase) | 12.17 (5.08) | 13.01 (5.09) | 13.94 (4.67) | 13.37 (4.69) | 13.36 (4.83)
  Week 12: Change from baseline (Bone Specific Alkaline Phosphatase): number analyzed (Participants) | 43 | 29 | 16 | 46 | 42
  Week 12: Change from baseline (Bone Specific Alkaline Phosphatase) | 0.48 (2.22) | 0.34 (4.24) | -0.68 (3.36) | -0.43 (2.50) | -0.11 (2.73)
  Week 16: Change from baseline (Bone Specific Alkaline Phosphatase): number analyzed (Participants) | 41 | 29 | 16 | 47 | 45
  Week 16: Change from baseline (Bone Specific Alkaline Phosphatase) | 0.86 (3.57) | 1.22 (7.58) | -1.18 (2.49) | 0.84 (3.55) | 0.48 (2.98)
  Baseline (Procollagen 1 N-Terminal Propeptide): number analyzed (Participants) | 47 | 30 | 17 | 50 | 52
  Baseline (Procollagen 1 N-Terminal Propeptide) | 58.1 (23.3) | 68.0 (24.7) | 67.6 (15.6) | 68.6 (29.3) | 59.5 (23.6)
  Week 12: Change from baseline (Procollagen 1 N-Terminal Propeptide): number analyzed (Participants) | 43 | 29 | 16 | 49 | 42
  Week 12: Change from baseline (Procollagen 1 N-Terminal Propeptide) | 5.0 (14.5) | 0.5 (10.9) | -5.7 (15.9) | -2.1 (13.7) | -0.7 (10.9)
  Week 16: Change from baseline (Procollagen 1 N-Terminal Propeptide): number analyzed (Participants) | 41 | 29 | 16 | 48 | 45
  Week 16: Change from baseline (Procollagen 1 N-Terminal Propeptide) | 3.6 (20.2) | -1.9 (9.7) | -0.9 (19.6) | -2.5 (15.4) | 0.0 (11.7)

52. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 in Clinical Laboratory Parameters Urinalysis: pH
Description: Urine for urinalysis was collected and sent to the central laboratory for analysis. Urine pH was measured on a pH scale.
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
pH
  Baseline (pH): number analyzed (Participants) | 47 | 31 | 17 | 51 | 52
  Baseline (pH) | 6.00 (0.83) | 6.10 (0.89) | 6.09 (0.92) | 6.21 (0.75) | 6.08 (0.72)
  Week 2: Change from baseline (pH): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (pH) | 0.10 (0.70) | 0.26 (0.90) | -0.15 (0.95) | -0.30 (0.83) | -0.20 (0.83)
  Week 4: Change from baseline (pH): number analyzed (Participants) | 45 | 31 | 17 | 50 | 48
  Week 4: Change from baseline (pH) | -0.11 (0.85) | 0.18 (1.31) | -0.09 (0.80) | -0.25 (0.83) | -0.09 (0.89)
  Week 12: Change from baseline (pH): number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (pH) | -0.05 (0.89) | 0.18 (1.06) | -0.19 (0.83) | -0.21 (0.78) | -0.06 (0.79)
  Week 16: Change from baseline (pH): number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16: Change from baseline (pH) | 0.05 (1.13) | 0.00 (1.12) | -0.03 (0.90) | -0.19 (0.84) | 0.07 (1.04)

53. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 in Clinical Laboratory Parameters Urinalysis: Specific Gravity
Description: Urine for urinalysis was collected and sent to the central laboratory for analysis.
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Unitless
  Baseline (Specific Gravity): number analyzed (Participants) | 47 | 31 | 17 | 51 | 52
  Baseline (Specific Gravity) | 1.0167 (0.0063) | 1.0167 (0.0083) | 1.0166 (0.0063) | 1.0154 (0.0064) | 1.0171 (0.0084)
  Week 2: Change from baseline (Specific Gravity): number analyzed (Participants) | 44 | 31 | 17 | 51 | 51
  Week 2: Change from baseline (Specific Gravity) | -0.0002 (0.0066) | -0.0011 (0.0085) | 0.0001 (0.0060) | 0.0005 (0.0068) | -0.0006 (0.0060)
  Week 4: Change from baseline (Specific Gravity): number analyzed (Participants) | 45 | 31 | 17 | 50 | 48
  Week 4: Change from baseline (Specific Gravity) | -0.0008 (0.0078) | 0.0012 (0.0086) | -0.0026 (0.0063) | 0.0015 (0.0067) | 0.0003 (0.0079)
  Week 12: Change from baseline (Specific Gravity): number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12: Change from baseline (Specific Gravity) | 0.0020 (0.0068) | 0.0015 (0.0102) | -0.0012 (0.0060) | 0.0002 (0.0068) | 0.0011 (0.0072)
  Week 16: Change from baseline (Specific Gravity): number analyzed (Participants) | 41 | 30 | 16 | 50 | 44
  Week 16: Change from baseline (Specific Gravity) | 0.0009 (0.0088) | 0.0002 (0.0093) | -0.0011 (0.0059) | 0.0020 (0.0066) | -0.0006 (0.0066)

54. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 in Clinical Laboratory Parameters Urinalysis: Glucose, Bilirubin, Ketones, Occult Blood, Protein, Urobilinogen and Nitrite
Description: Urine for urinalysis was collected and sent to the central laboratory for analysis. Clinical relevance was judged by the investigator. Assessment was done using standard laboratory practice.
  For evaluation of the chemical properties of the urine sample test strips were used which have test pads of chemicals that change color when they come in contact with reagents. The degree of color change correlates with the amount of reagent present. Each color block represents a range of values. Range and direction of scores for reagents nitrite and urobilinogen: negative = normal; positive = abnormal. Range and direction of scores for all other reagents tested: negative = normal; trace, 1+, 2+, 3+ = abnormal, the higher the value, the higher the concentration of the reagent tested.
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 47 | 31 | 17 | 52 | 52
Participants
  Baseline (Glucose): Negative: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Glucose): Negative | 46 | 30 | 17 | 49 | 48
  Baseline (Glucose): Trace | 1 | 0 | 0 | 0 | 1
  Baseline (Glucose): 1+ | 0 | 1 | 0 | 0 | 0
  Baseline (Glucose): 2+ | 0 | 0 | 0 | 0 | 0
  Baseline (Glucose): 3+ | 0 | 0 | 0 | 0 | 2
  Week 2 (Glucose): Negative: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Glucose): Negative | 44 | 31 | 17 | 52 | 49
  Week 2 (Glucose): Trace: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Glucose): Trace | 0 | 0 | 0 | 0 | 0
  Week 2 (Glucose): 1+: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Glucose): 1+ | 0 | 0 | 0 | 0 | 1
  Week 2 (Glucose): 2+: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Glucose): 2+ | 0 | 0 | 0 | 0 | 0
  Week 2 (Glucose): 3+: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Glucose): 3+ | 0 | 0 | 0 | 0 | 1
  Week 4 (Glucose): Negative: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Glucose): Negative | 45 | 30 | 17 | 51 | 46
  Week 4 (Glucose): Trace: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Glucose): Trace | 0 | 1 | 0 | 0 | 0
  Week 4 (Glucose): 1+: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Glucose): 1+ | 0 | 0 | 0 | 0 | 0
  Week 4 (Glucose): 2+: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Glucose): 2+ | 0 | 0 | 0 | 0 | 0
  Week 4 (Glucose): 3+: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Glucose): 3+ | 0 | 0 | 0 | 0 | 2
  Week 12 (Glucose): Negative: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Glucose): Negative | 43 | 30 | 16 | 47 | 40
  Week 12 (Glucose): Trace: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Glucose): Trace | 0 | 0 | 0 | 1 | 1
  Week 12 (Glucose): 1+: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Glucose): 1+ | 0 | 0 | 0 | 0 | 1
  Week 12 (Glucose): 2+: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Glucose): 2+ | 0 | 0 | 0 | 0 | 0
  Week 12 (Glucose): 3+: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Glucose): 3+ | 0 | 0 | 0 | 1 | 2
  Week 16 (Glucose): Negative: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Glucose): Negative | 40 | 29 | 16 | 50 | 43
  Week 16 (Glucose): Trace: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Glucose): Trace | 0 | 1 | 0 | 0 | 0
  Week 16 (Glucose): 1+: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Glucose): 1+ | 1 | 0 | 0 | 0 | 0
  Week 16 (Glucose): 2+: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Glucose): 2+ | 0 | 0 | 0 | 0 | 0
  Week 16 (Glucose): 3+: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Glucose): 3+ | 0 | 0 | 0 | 1 | 1
  Baseline (Bilirubin): Negative: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Bilirubin): Negative | 47 | 31 | 17 | 49 | 51
  Baseline (Bilirubin): 1+: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Bilirubin): 1+ | 0 | 0 | 0 | 0 | 0
  Week 2 (Bilirubin): Negative: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Bilirubin): Negative | 44 | 31 | 17 | 52 | 51
  Week 2 (Bilirubin): 1+: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Bilirubin): 1+ | 0 | 0 | 0 | 0 | 0
  Week 4 (Bilirubin): Negative: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Bilirubin): Negative | 45 | 31 | 17 | 51 | 48
  Week 4 (Bilirubin): 1+: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Bilirubin): 1+ | 0 | 0 | 0 | 0 | 0
  Week 12 (Bilirubin): Negative: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Bilirubin): Negative | 43 | 30 | 16 | 49 | 44
  Week 12 (Bilirubin): 1+: number analyzed (Participants) | 43 | 30 | 16 | 52 | 44
  Week 12 (Bilirubin): 1+ | 0 | 0 | 0 | 0 | 0
  Week 16 (Bilirubin): Negative: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Bilirubin): Negative | 41 | 29 | 16 | 51 | 44
  Week 16 (Bilirubin): 1+: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Bilirubin): 1+ | 0 | 1 | 0 | 0 | 0
  Baseline (Ketones): Negative: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Ketones): Negative | 46 | 31 | 17 | 48 | 50
  Baseline (Ketones): Trace: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Ketones): Trace | 1 | 0 | 0 | 1 | 1
  Week 2 (Ketones): Negative: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Ketones): Negative | 44 | 31 | 17 | 51 | 50
  Week 2 (Ketones): Trace: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Ketones): Trace | 0 | 0 | 0 | 1 | 1
  Week 4 (Ketones): Negative: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Ketones): Negative | 45 | 31 | 17 | 50 | 48
  Week 4 (Ketones): Trace: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Ketones): Trace | 0 | 0 | 0 | 1 | 0
  Week 12 (Ketones): Negative: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Ketones): Negative | 42 | 30 | 16 | 48 | 43
  Week 12 (Ketones): Trace: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Ketones): Trace | 1 | 0 | 0 | 1 | 1
  Week 16 (Ketones): Negative: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Ketones): Negative | 41 | 30 | 16 | 50 | 44
  Week 16 (Ketones): Trace: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Ketones): Trace | 0 | 0 | 0 | 1 | 0
  Baseline (Occult Blood): Negative: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Occult Blood): Negative | 46 | 28 | 15 | 42 | 47
  Baseline (Occult Blood): Trace: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Occult Blood): Trace | 0 | 3 | 1 | 3 | 4
  Baseline (Occult Blood): 1+: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Occult Blood): 1+ | 1 | 0 | 0 | 3 | 0
  Baseline (Occult Blood): 2+: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Occult Blood): 2+ | 0 | 0 | 0 | 1 | 0
  Baseline (Occult Blood): 3+: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Occult Blood): 3+ | 0 | 0 | 1 | 0 | 0
  Week 2 (Occult Blood): Negative: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Occult Blood): Negative | 42 | 29 | 17 | 45 | 47
  Week 2 (Occult Blood): Trace: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Occult Blood): Trace | 1 | 2 | 0 | 1 | 3
  Week 2 (Occult Blood): 1+: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Occult Blood): 1+ | 1 | 0 | 0 | 5 | 1
  Week 2 (Occult Blood): 2+: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Occult Blood): 2+ | 0 | 0 | 0 | 1 | 0
  Week 2 (Occult Blood): 3+: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Occult Blood): 3+ | 0 | 0 | 0 | 0 | 0
  Week 4 (Occult Blood): Negative: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Occult Blood): Negative | 43 | 28 | 17 | 42 | 47
  Week 4 (Occult Blood): Trace: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Occult Blood): Trace | 2 | 1 | 0 | 5 | 1
  Week 4 (Occult Blood): 1+: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Occult Blood): 1+ | 0 | 2 | 0 | 3 | 0
  Week 4 (Occult Blood): 2+: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Occult Blood): 2+ | 0 | 0 | 0 | 0 | 0
  Week 4 (Occult Blood): 3+: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Occult Blood): 3+ | 0 | 0 | 0 | 1 | 0
  Week 12 (Occult Blood): Negative: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Occult Blood): Negative | 40 | 30 | 13 | 40 | 42
  Week 12 (Occult Blood): Trace: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Occult Blood): Trace | 1 | 0 | 1 | 5 | 2
  Week 12 (Occult Blood): 1+: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Occult Blood): 1+ | 2 | 0 | 1 | 3 | 0
  Week 12 (Occult Blood): 2+: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Occult Blood): 2+ | 0 | 0 | 1 | 1 | 0
  Week 12 (Occult Blood): 3+: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Occult Blood): 3+ | 0 | 0 | 0 | 0 | 0
  Week 16 (Occult Blood): Negative: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Occult Blood): Negative | 38 | 27 | 14 | 45 | 39
  Week 16 (Occult Blood): Trace: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Occult Blood): Trace | 2 | 3 | 1 | 3 | 4
  Week 16 (Occult Blood): 1+: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Occult Blood): 1+ | 0 | 0 | 0 | 3 | 1
  Week 16 (Occult Blood): 2+: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Occult Blood): 2+ | 1 | 0 | 0 | 0 | 0
  Week 16 (Occult Blood): 3+: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Occult Blood): 3+ | 0 | 0 | 1 | 0 | 0
  Baseline (Protein): Negative: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Protein): Negative | 45 | 31 | 16 | 48 | 49
  Baseline (Protein): Trace: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Protein): Trace | 2 | 0 | 1 | 1 | 1
  Baseline (Protein): 1+: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Protein): 1+ | 0 | 0 | 0 | 0 | 1
  Baseline (Protein): 2+: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Protein): 2+ | 0 | 0 | 0 | 0 | 0
  Baseline (Protein): 3+: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Protein): 3+ | 0 | 0 | 0 | 0 | 0
  Week 2 (Protein): Negative: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Protein): Negative | 44 | 31 | 17 | 52 | 49
  Week 2 (Protein): Trace: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Protein): Trace | 0 | 0 | 0 | 0 | 0
  Week 2 (Protein): 1+: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Protein): 1+ | 0 | 0 | 0 | 0 | 0
  Week 2 (Protein): 2+: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Protein): 2+ | 0 | 0 | 0 | 0 | 2
  Week 2 (Protein): 3+: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Protein): 3+ | 0 | 0 | 0 | 0 | 0
  Week 4 (Protein): Negative: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Protein): Negative | 44 | 31 | 17 | 49 | 45
  Week 4 (Protein): Trace: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Protein): Trace | 0 | 0 | 0 | 2 | 3
  Week 4 (Protein): 1+: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Protein): 1+ | 1 | 0 | 0 | 0 | 0
  Week 4 (Protein): 2+: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Protein): 2+ | 0 | 0 | 0 | 0 | 0
  Week 4 (Protein): 3+: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Protein): 3+ | 0 | 0 | 0 | 0 | 0
  Week 12 (Protein): Negative: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Protein): Negative | 41 | 30 | 14 | 47 | 43
  Week 12 (Protein): Trace: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Protein): Trace | 1 | 0 | 0 | 1 | 1
  Week 12 (Protein): 1+: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Protein): 1+ | 1 | 0 | 2 | 1 | 0
  Week 12 (Protein): 2+: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Protein): 2+ | 0 | 0 | 0 | 0 | 0
  Week 12 (Protein): 3+: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Protein): 3+ | 0 | 0 | 0 | 0 | 0
  Week 16 (Protein): Negative: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Protein): Negative | 39 | 30 | 15 | 50 | 43
  Week 16 (Protein): Trace: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Protein): Trace | 1 | 0 | 0 | 0 | 1
  Week 16 (Protein): 1+: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Protein): 1+ | 0 | 0 | 0 | 1 | 0
  Week 16 (Protein): 2+: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Protein): 2+ | 0 | 0 | 1 | 0 | 0
  Week 16 (Protein): 3+: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Protein): 3+ | 1 | 0 | 0 | 0 | 0
  Baseline (Urobilinogen): Negative: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Urobilinogen): Negative | 47 | 31 | 17 | 49 | 51
  Week 2 (Urobilinogen): Negative: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Urobilinogen): Negative | 44 | 31 | 17 | 52 | 51
  Week 4 (Urobilinogen): Negative: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Urobilinogen): Negative | 45 | 31 | 17 | 51 | 48
  Week 12 (Urobilinogen): Negative: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Urobilinogen): Negative | 43 | 30 | 16 | 49 | 44
  Week 16 (Urobilinogen): Negative: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Urobilinogen): Negative | 41 | 30 | 16 | 51 | 44
  Baseline (Nitrite): Negative: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Nitrite): Negative | 47 | 29 | 17 | 48 | 48
  Baseline (Nitrite): Positive: number analyzed (Participants) | 47 | 31 | 17 | 49 | 51
  Baseline (Nitrite): Positive | 0 | 2 | 0 | 1 | 3
  Week 2 (Nitrite): Negative: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Nitrite): Negative | 44 | 29 | 17 | 51 | 47
  Week 2 (Nitrite): Positive: number analyzed (Participants) | 44 | 31 | 17 | 52 | 51
  Week 2 (Nitrite): Positive | 0 | 2 | 0 | 1 | 4
  Week 4 (Nitrite): Negative: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Nitrite): Negative | 45 | 29 | 17 | 50 | 47
  Week 4 (Nitrite): Positive: number analyzed (Participants) | 45 | 31 | 17 | 51 | 48
  Week 4 (Nitrite): Positive | 0 | 2 | 0 | 1 | 1
  Week 12 (Nitrite): Negative: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Nitrite): Negative | 42 | 29 | 16 | 49 | 42
  Week 12 (Nitrite): Positive: number analyzed (Participants) | 43 | 30 | 16 | 49 | 44
  Week 12 (Nitrite): Positive | 1 | 1 | 0 | 0 | 2
  Week 16 (Nitrite): Negative: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Nitrite): Negative | 41 | 30 | 16 | 51 | 42
  Week 16 (Nitrite): Positive: number analyzed (Participants) | 41 | 30 | 16 | 51 | 44
  Week 16 (Nitrite): Positive | 0 | 0 | 0 | 0 | 2

55. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 in Clinical Laboratory Parameters Urinalysis: Erythrocytes and Leukocytes
Description: Urine for urinalysis was collected and sent to the central laboratory for analysis. Results are reported according to the amount present in the microscope's field of view at high magnification (/HPF [high-power field]).
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: Participants in safety analysis set (SAF) with evaluable data at baseline and each week were reported. Only some participants have baseline or post baseline value for this endpoint therefore the numbers are much lower than expected.
Measure: Mean (Standard Deviation); unit: cells/HPF
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 18 | 12 | 7 | 23 | 23
cells/HPF
  Baseline (Erythrocytes (/HPF)) | 1.3 (1.5) | 0.8 (1.1) | 2.0 (2.6) | 1.5 (2.4) | 0.6 (0.7)
  Week 2: Change from baseline (Erythrocytes (/HPF)): number analyzed (Participants) | 7 | 5 | 2 | 9 | 14
  Week 2: Change from baseline (Erythrocytes (/HPF)) | -0.6 (2.6) | -0.6 (0.5) | -1.0 (1.4) | -0.8 (4.0) | 0.9 (3.0)
  Week 4: Change from baseline (Erythrocytes (/HPF)): number analyzed (Participants) | 9 | 4 | 3 | 13 | 9
  Week 4: Change from baseline (Erythrocytes (/HPF)) | -0.1 (1.6) | 0.5 (1.3) | -2.7 (3.1) | -0.5 (3.1) | 0.3 (1.1)
  Week 12: Change from baseline (Erythrocytes (/HPF)): number analyzed (Participants) | 8 | 7 | 5 | 11 | 11
  Week 12: Change from baseline (Erythrocytes (/HPF)) | -0.4 (2.2) | -0.4 (0.8) | 0.4 (0.5) | 1.4 (3.7) | 0.2 (1.5)
  Week 16: Change from baseline (Erythrocytes (/HPF)): number analyzed (Participants) | 10 | 3 | 4 | 8 | 9
  Week 16: Change from baseline (Erythrocytes (/HPF)) | -0.3 (2.1) | -0.7 (1.2) | -1.5 (2.4) | 0.3 (2.1) | 0.1 (0.3)
  Baseline (Leukocytes (/HPF)): number analyzed (Participants) | 18 | 12 | 7 | 22 | 23
  Baseline (Leukocytes (/HPF)) | 9.5 (16.2) | 2.6 (4.3) | 1.6 (1.7) | 5.3 (11.9) | 3.0 (5.8)
  Week 2: Change from baseline (Leukocytes (/HPF)): number analyzed (Participants) | 7 | 5 | 2 | 8 | 14
  Week 2: Change from baseline (Leukocytes (/HPF)) | -6.7 (15.9) | 0.0 (3.6) | 0.5 (2.1) | -1.0 (2.7) | -0.4 (6.4)
  Week 4: Change from baseline (Leukocytes (/HPF)): number analyzed (Participants) | 9 | 3 | 3 | 12 | 9
  Week 4: Change from baseline (Leukocytes (/HPF)) | -6.0 (20.9) | 1.0 (1.0) | 6.3 (11.8) | 0.3 (4.1) | 0.8 (5.8)
  Week 12: Change from baseline (Leukocytes (/HPF)): number analyzed (Participants) | 8 | 6 | 5 | 10 | 11
  Week 12: Change from baseline (Leukocytes (/HPF)) | 6.4 (47.9) | 3.5 (6.7) | 0.6 (3.0) | 0.6 (2.3) | -1.5 (5.1)
  Week 16: Change from baseline (Leukocytes (/HPF)): number analyzed (Participants) | 10 | 3 | 4 | 8 | 9
  Week 16: Change from baseline (Leukocytes (/HPF)) | -7.6 (21.9) | 3.0 (4.4) | 3.0 (4.2) | 0.6 (1.3) | 13.3 (33.4)

56. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 in Clinical Laboratory Parameters Urinalysis: Hyaline Casts
Description: Urine for urinalysis was collected and sent to the central laboratory for analysis. Results are reported according to the amount present in the microscope's field of view at low magnification (/LPF [low-power field]).
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: cells/LPF
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 18 | 12 | 7 | 23 | 23
cells/LPF
  Baseline (Hyaline Casts (/LPF) | 1.9 (2.0) | 0.8 (1.6) | 0.1 (0.4) | 0.8 (1.4) | 1.7 (6.2)
  Week 2: Change from baseline (Hyaline Casts (/LPF)): number analyzed (Participants) | 7 | 5 | 2 | 9 | 14
  Week 2: Change from baseline (Hyaline Casts (/LPF)) | -1.1 (2.7) | -0.6 (1.5) | 0.0 (0.0) | -0.1 (0.6) | 0.1 (1.5)
  Week 4: Change from baseline (Hyaline Casts (/LPF)): number analyzed (Participants) | 9 | 4 | 3 | 13 | 9
  Week 4: Change from baseline (Hyaline Casts (/LPF)) | -0.2 (3.6) | -0.5 (1.0) | 5.3 (6.8) | 0.3 (1.8) | -0.4 (1.7)
  Week 12: Change from baseline (Hyaline Casts (/LPF)): number analyzed (Participants) | 8 | 7 | 5 | 11 | 11
  Week 12: Change from baseline (Hyaline Casts (/LPF)) | -0.3 (2.8) | -0.1 (1.5) | 2.2 (4.4) | -0.3 (0.8) | -2.8 (9.0)
  Week 16: Change from baseline (Hyaline Casts (/LPF)): number analyzed (Participants) | 10 | 3 | 4 | 8 | 9
  Week 16: Change from baseline (Hyaline Casts (/LPF)) | -1.2 (2.9) | 0.7 (1.2) | 0.5 (1.0) | 0.1 (0.8) | -0.2 (0.8)

57. Secondary Outcome: Change From Baseline at Weeks 2, 4, 12 and 16 in Clinical Laboratory Parameters Urinalysis: Bacteria, Yeast Cells, Granular Casts, RBC Casts, Waxy Casts, WBC Casts, Calcium Oxalate Crystals, Triple Phosphate Crystals and Uric Acid Crystals
Description: Urine for urinalysis was collected and sent to the central laboratory for analysis. The evaluation of components in the urine samples such as bacteria, yeast, red blood cells (RBC), white blood cells (WBC), casts and crystals was performed by microscopy. Results are reported according to the amount present in the microscope's field of view at low magnification (/LPF [low-power field]) and high magnification (/HPF [high-power field]).
  Range and direction of scores microscopic identification of urine components:
  * Bacteria: none seen, 1+, 2+, 3+,4+, TNTC (too numerous to count).
  * Other urine components: none seen=normal; few, moderate, many, TNTC = abnormal. The higher the value, the higher the concentration of the component evaluated.
Time Frame: From baseline to Weeks 2, 4, 12 and 16
Population: as for outcome 55
Measure: Number; unit: Participants
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
Number analyzed (Participants) | 13 | 11 | 8 | 18 | 19
Participants
  Baseline (Bacteria(/HPF)): None seen: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Bacteria(/HPF)): None seen | 4 | 4 | 2 | 9 | 7
  Baseline (Bacteria(/HPF)): 1+: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Bacteria(/HPF)): 1+ | 4 | 3 | 1 | 6 | 5
  Baseline (Bacteria(/HPF)): 2+: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Bacteria(/HPF)): 2+ | 0 | 1 | 1 | 1 | 2
  Baseline (Bacteria(/HPF)): 3+: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Bacteria(/HPF)): 3+ | 0 | 1 | 0 | 0 | 2
  Baseline (Bacteria(/HPF)): 4+: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Bacteria(/HPF)): 4+ | 0 | 0 | 1 | 1 | 1
  Baseline (Bacteria(/HPF)): TNTC: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Bacteria(/HPF)): TNTC | 1 | 2 | 0 | 0 | 2
  Week 2 (Bacteria(/HPF)): None seen: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Bacteria(/HPF)): None seen | 3 | 3 | 1 | 5 | 6
  Week 2 (Bacteria(/HPF)): 1+: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Bacteria(/HPF)): 1+ | 1 | 2 | 1 | 4 | 4
  Week 2 (Bacteria(/HPF)): 2+: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Bacteria(/HPF)): 2+ | 1 | 2 | 1 | 0 | 6
  Week 2 (Bacteria(/HPF)): 3+: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Bacteria(/HPF)): 3+ | 0 | 1 | 0 | 1 | 1
  Week 2 (Bacteria(/HPF)): 4+: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Bacteria(/HPF)): 4+ | 2 | 0 | 0 | 0 | 0
  Week 2 (Bacteria(/HPF)): TNTC: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Bacteria(/HPF)): TNTC | 1 | 1 | 0 | 1 | 1
  Week 4 (Bacteria(/HPF)): None seen: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Bacteria(/HPF)): None seen | 7 | 3 | 1 | 9 | 2
  Week 4 (Bacteria(/HPF)): 1+: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Bacteria(/HPF)): 1+ | 0 | 0 | 1 | 1 | 3
  Week 4 (Bacteria(/HPF)): 2+: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Bacteria(/HPF)): 2+ | 2 | 0 | 1 | 4 | 3
  Week 4 (Bacteria(/HPF)): 3+: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Bacteria(/HPF)): 3+ | 0 | 0 | 0 | 0 | 1
  Week 4 (Bacteria(/HPF)): 4+: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Bacteria(/HPF)): 4+ | 0 | 0 | 0 | 0 | 2
  Week 4 (Bacteria(/HPF)): TNTC: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Bacteria(/HPF)): TNTC | 2 | 3 | 0 | 1 | 2
  Week 12 (Bacteria(/HPF)): None seen: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Bacteria(/HPF)): None seen | 1 | 3 | 3 | 11 | 3
  Week 12 (Bacteria(/HPF)): 1+: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Bacteria(/HPF)): 1+ | 7 | 2 | 3 | 3 | 3
  Week 12 (Bacteria(/HPF)): 2+: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Bacteria(/HPF)): 2+ | 1 | 0 | 2 | 3 | 5
  Week 12 (Bacteria(/HPF)): 3+: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Bacteria(/HPF)): 3+ | 1 | 0 | 0 | 1 | 0
  Week 12 (Bacteria(/HPF)): 4+: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Bacteria(/HPF)): 4+ | 0 | 1 | 0 | 0 | 0
  Week 12 (Bacteria(/HPF)): TNTC: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Bacteria(/HPF)): TNTC | 2 | 2 | 0 | 0 | 1
  Week 16 (Bacteria(/HPF)): None seen: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Bacteria(/HPF)): None seen | 2 | 3 | 2 | 6 | 4
  Week 16 (Bacteria(/HPF)): 1+: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Bacteria(/HPF)): 1+ | 5 | 0 | 0 | 3 | 3
  Week 16 (Bacteria(/HPF)): 2+: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Bacteria(/HPF)): 2+ | 4 | 2 | 1 | 1 | 1
  Week 16 (Bacteria(/HPF)): 3+: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Bacteria(/HPF)): 3+ | 1 | 0 | 0 | 1 | 2
  Week 16 (Bacteria(/HPF)): 4+: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Bacteria(/HPF)): 4+ | 1 | 1 | 2 | 0 | 3
  Week 16 (Bacteria(/HPF)): TNTC: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Bacteria(/HPF)): TNTC | 0 | 0 | 0 | 1 | 1
  Baseline (Yeast Cells(/HPF)): None seen: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Yeast Cells(/HPF)): None seen | 9 | 11 | 5 | 17 | 19
  Baseline (Yeast Cells(/HPF)): Few: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Yeast Cells(/HPF)): Few | 0 | 0 | 0 | 0 | 0
  Week 2 (Yeast Cells(/HPF)): None seen: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Yeast Cells(/HPF)): None seen | 8 | 9 | 3 | 11 | 17
  Week 2 (Yeast Cells(/HPF)): Few: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Yeast Cells(/HPF)): Few | 0 | 0 | 0 | 0 | 1
  Week 4 (Yeast Cells(/HPF)): None seen: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Yeast Cells(/HPF)): None seen | 11 | 6 | 3 | 15 | 13
  Week 4 (Yeast Cells(/HPF)): Few: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Yeast Cells(/HPF)): Few | 0 | 0 | 0 | 0 | 0
  Week 12 (Yeast Cells(/HPF)): None seen: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Yeast Cells(/HPF)): None seen | 12 | 8 | 8 | 18 | 12
  Week 12 (Yeast Cells(/HPF)): Few: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Yeast Cells(/HPF)): Few | 0 | 0 | 0 | 0 | 0
  Week 16 (Yeast Cells(/HPF)): None seen: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Yeast Cells(/HPF)): None seen | 13 | 6 | 5 | 12 | 14
  Week 16 (Yeast Cells(/HPF)): Few: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Yeast Cells(/HPF)): Few | 0 | 0 | 0 | 0 | 0
  Baseline (Granular Casts(/LPF)): None seen: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Granular Casts(/LPF)): None seen | 9 | 11 | 5 | 17 | 19
  Week 2: (Granular Casts(/LPF)): None seen: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2: (Granular Casts(/LPF)): None seen | 8 | 9 | 3 | 11 | 18
  Week 4: (Granular Casts(/LPF)): None seen: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4: (Granular Casts(/LPF)): None seen | 11 | 6 | 3 | 15 | 13
  Week 12: (Granular Casts(/LPF)): None seen: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12: (Granular Casts(/LPF)): None seen | 12 | 8 | 8 | 18 | 12
  Week 16: (Granular Casts(/LPF)): None seen: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16: (Granular Casts(/LPF)): None seen | 13 | 6 | 5 | 12 | 14
  Baseline (RBC Casts(/LPF)): None seen: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (RBC Casts(/LPF)): None seen | 9 | 11 | 5 | 17 | 19
  Week 2 (RBC Casts(/LPF)): None seen: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (RBC Casts(/LPF)): None seen | 8 | 9 | 3 | 11 | 18
  Week 4 (RBC Casts(/LPF)): None seen: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (RBC Casts(/LPF)): None seen | 11 | 6 | 3 | 15 | 13
  Week 12 (RBC Casts(/LPF)): None seen: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (RBC Casts(/LPF)): None seen | 12 | 8 | 8 | 18 | 12
  Week 16 (RBC Casts(/LPF)): None seen: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (RBC Casts(/LPF)): None seen | 13 | 6 | 5 | 12 | 14
  Baseline (Waxy Casts(/LPF)): None seen: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Waxy Casts(/LPF)): None seen | 9 | 11 | 5 | 17 | 19
  Week 2 (Waxy Casts(/LPF)): None seen: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Waxy Casts(/LPF)): None seen | 8 | 9 | 3 | 11 | 18
  Week 4 (Waxy Casts(/LPF)): None seen: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Waxy Casts(/LPF)): None seen | 11 | 6 | 3 | 15 | 13
  Week 12 (Waxy Casts(/LPF)): None seen: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Waxy Casts(/LPF)): None seen | 12 | 8 | 8 | 18 | 12
  Week 16 (Waxy Casts(/LPF)): None seen: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Waxy Casts(/LPF)): None seen | 13 | 6 | 5 | 12 | 14
  Baseline (WBC Casts(/LPF)): None seen: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (WBC Casts(/LPF)): None seen | 9 | 11 | 5 | 17 | 19
  Week 2 (WBC Casts(/LPF)): None seen: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (WBC Casts(/LPF)): None seen | 8 | 9 | 3 | 11 | 18
  Week 4 (WBC Casts(/LPF)): None seen: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (WBC Casts(/LPF)): None seen | 11 | 6 | 3 | 15 | 13
  Week 12 (WBC Casts(/LPF)): None seen: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (WBC Casts(/LPF)): None seen | 12 | 8 | 8 | 18 | 12
  Week 16 (WBC Casts(/LPF)): None seen: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (WBC Casts(/LPF)): None seen | 13 | 6 | 5 | 12 | 14
  Baseline (Calcium Oxalate Crystals(/HPF)): None seen: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Calcium Oxalate Crystals(/HPF)): None seen | 8 | 11 | 5 | 13 | 16
  Baseline (Calcium Oxalate Crystals(/HPF)): Few: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Calcium Oxalate Crystals(/HPF)): Few | 1 | 0 | 0 | 2 | 2
  Baseline (Calcium Oxalate Crystals(/HPF)): Moderate: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Calcium Oxalate Crystals(/HPF)): Moderate | 0 | 0 | 0 | 0 | 1
  Baseline (Calcium Oxalate Crystals(/HPF)): Many: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Calcium Oxalate Crystals(/HPF)): Many | 0 | 0 | 0 | 2 | 0
  Baseline (Calcium Oxalate Crystals(/HPF)): TNTC: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Calcium Oxalate Crystals(/HPF)): TNTC | 0 | 0 | 0 | 0 | 0
  Week 2 (Calcium Oxalate Crystals(/HPF)): None seen: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Calcium Oxalate Crystals(/HPF)): None seen | 6 | 8 | 3 | 9 | 17
  Week 2 (Calcium Oxalate Crystals(/HPF)): Few: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Calcium Oxalate Crystals(/HPF)): Few | 2 | 0 | 0 | 1 | 0
  Week 2 (Calcium Oxalate Crystals(/HPF)): Moderate: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Calcium Oxalate Crystals(/HPF)): Moderate | 0 | 0 | 0 | 0 | 1
  Week 2 (Calcium Oxalate Crystals(/HPF)): Many: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Calcium Oxalate Crystals(/HPF)): Many | 0 | 1 | 0 | 1 | 0
  Week 2 (Calcium Oxalate Crystals(/HPF)): TNTC: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Calcium Oxalate Crystals(/HPF)): TNTC | 0 | 0 | 0 | 0 | 0
  Week 4 (Calcium Oxalate Crystals(/HPF)): None seen: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Calcium Oxalate Crystals(/HPF)): None seen | 9 | 5 | 3 | 12 | 10
  Week 4 (Calcium Oxalate Crystals(/HPF)): Few: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Calcium Oxalate Crystals(/HPF)): Few | 0 | 0 | 0 | 1 | 1
  Week 4 (Calcium Oxalate Crystals(/HPF)): Moderate: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Calcium Oxalate Crystals(/HPF)): Moderate | 1 | 1 | 0 | 1 | 0
  Week 4 (Calcium Oxalate Crystals(/HPF)): Many: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Calcium Oxalate Crystals(/HPF)): Many | 1 | 0 | 0 | 1 | 1
  Week 4 (Calcium Oxalate Crystals(/HPF)): TNTC: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Calcium Oxalate Crystals(/HPF)): TNTC | 0 | 0 | 0 | 0 | 1
  Week 12 (Calcium Oxalate Crystals(/HPF)): None seen: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Calcium Oxalate Crystals(/HPF)): None seen | 11 | 7 | 8 | 16 | 11
  Week 12 (Calcium Oxalate Crystals(/HPF)): Few: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Calcium Oxalate Crystals(/HPF)): Few | 1 | 0 | 0 | 0 | 1
  Week 12 (Calcium Oxalate Crystals(/HPF)): Moderate: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Calcium Oxalate Crystals(/HPF)): Moderate | 0 | 1 | 0 | 1 | 0
  Week 12 (Calcium Oxalate Crystals(/HPF)): Many: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Calcium Oxalate Crystals(/HPF)): Many | 0 | 0 | 0 | 1 | 0
  Week 12 (Calcium Oxalate Crystals(/HPF)): TNTC: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Calcium Oxalate Crystals(/HPF)): TNTC | 0 | 0 | 0 | 0 | 0
  Week 16 (Calcium Oxalate Crystals(/HPF)): None seen: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Calcium Oxalate Crystals(/HPF)): None seen | 10 | 4 | 5 | 11 | 14
  Week 16 (Calcium Oxalate Crystals(/HPF)): Few: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Calcium Oxalate Crystals(/HPF)): Few | 2 | 2 | 0 | 0 | 0
  Week 16 (Calcium Oxalate Crystals(/HPF)): Moderate: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Calcium Oxalate Crystals(/HPF)): Moderate | 1 | 0 | 0 | 0 | 0
  Week 16 (Calcium Oxalate Crystals(/HPF)): Many: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Calcium Oxalate Crystals(/HPF)): Many | 0 | 0 | 0 | 1 | 0
  Week 16 (Calcium Oxalate Crystals(/HPF)): TNTC: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Calcium Oxalate Crystals(/HPF)): TNTC | 0 | 0 | 0 | 0 | 0
  Baseline (Triple Phosphate Crystals(/HPF)): None seen: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Triple Phosphate Crystals(/HPF)): None seen | 9 | 11 | 5 | 17 | 19
  Week 2 (Triple Phosphate Crystals(/HPF)): None seen: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Triple Phosphate Crystals(/HPF)): None seen | 8 | 9 | 3 | 11 | 18
  Week 4 (Triple Phosphate Crystals(/HPF)): None seen: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Triple Phosphate Crystals(/HPF)): None seen | 11 | 6 | 3 | 15 | 13
  Week 12 (Triple Phosphate Crystals(/HPF)): None seen: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Triple Phosphate Crystals(/HPF)): None seen | 12 | 8 | 8 | 18 | 12
  Week 16 (Triple Phosphate Crystals(/HPF)): None seen: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Triple Phosphate Crystals(/HPF)): None seen | 13 | 6 | 5 | 12 | 14
  Baseline (Uric Acid Crystals(/HPF)): None seen: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Uric Acid Crystals(/HPF)): None seen | 9 | 11 | 5 | 16 | 19
  Baseline (Uric Acid Crystals(/HPF)): Few: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Uric Acid Crystals(/HPF)): Few | 0 | 0 | 0 | 1 | 0
  Baseline (Uric Acid Crystals(/HPF)): Moderate: number analyzed (Participants) | 9 | 11 | 5 | 17 | 19
  Baseline (Uric Acid Crystals(/HPF)): Moderate | 0 | 0 | 0 | 0 | 0
  Week 2 (Uric Acid Crystals(/HPF)): None seen: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Uric Acid Crystals(/HPF)): None seen | 8 | 9 | 3 | 11 | 18
  Week 2 (Uric Acid Crystals(/HPF)): Few: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Uric Acid Crystals(/HPF)): Few | 0 | 0 | 0 | 0 | 0
  Week 2 (Uric Acid Crystals(/HPF)): Moderate: number analyzed (Participants) | 8 | 9 | 3 | 11 | 18
  Week 2 (Uric Acid Crystals(/HPF)): Moderate | 0 | 0 | 0 | 0 | 0
  Week 4 (Uric Acid Crystals(/HPF)): None seen: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Uric Acid Crystals(/HPF)): None seen | 11 | 6 | 3 | 14 | 12
  Week 4 (Uric Acid Crystals(/HPF)): Few: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Uric Acid Crystals(/HPF)): Few | 0 | 0 | 0 | 0 | 1
  Week 4 (Uric Acid Crystals(/HPF)): Moderate: number analyzed (Participants) | 11 | 6 | 3 | 15 | 13
  Week 4 (Uric Acid Crystals(/HPF)): Moderate | 0 | 0 | 0 | 1 | 0
  Week 12 (Uric Acid Crystals(/HPF)): None seen: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Uric Acid Crystals(/HPF)): None seen | 11 | 8 | 8 | 18 | 12
  Week 12 (Uric Acid Crystals(/HPF)): Few: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Uric Acid Crystals(/HPF)): Few | 1 | 0 | 0 | 0 | 0
  Week 12 (Uric Acid Crystals(/HPF)): Moderate: number analyzed (Participants) | 12 | 8 | 8 | 18 | 12
  Week 12 (Uric Acid Crystals(/HPF)): Moderate | 0 | 0 | 0 | 0 | 0
  Week 16 (Uric Acid Crystals(/HPF)): None seen: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Uric Acid Crystals(/HPF)): None seen | 13 | 6 | 4 | 11 | 14
  Week 16 (Uric Acid Crystals(/HPF)): Few: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Uric Acid Crystals(/HPF)): Few | 0 | 0 | 1 | 1 | 0
  Week 16 (Uric Acid Crystals(/HPF)): Moderate: number analyzed (Participants) | 13 | 6 | 5 | 12 | 14
  Week 16 (Uric Acid Crystals(/HPF)): Moderate | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: On or after first dosing with randomised study treatment up to Week 16. Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study, up to 1 year.
Arm/Group | Placebo | 40 mg Elinzanetant (BAY3427080) | 80 mg Elinzanetant (BAY3427080) | 120 mg Elinzanetant (BAY3427080) | 160 mg Elinzanetant (BAY3427080)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/31 | 0/17 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 2/47 | 0/31 | 1/17 | 1/52 | 1/52
Other Adverse Events (participants affected / at risk) | 18/47 | 13/31 | 14/17 | 23/52 | 23/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | 40 mg Elinzanetant (BAY3427080) (N=31) | 80 mg Elinzanetant (BAY3427080) (N=17) | 120 mg Elinzanetant (BAY3427080) (N=52) | 160 mg Elinzanetant (BAY3427080) (N=52)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | 40 mg Elinzanetant (BAY3427080) (N=31) | 80 mg Elinzanetant (BAY3427080) (N=17) | 120 mg Elinzanetant (BAY3427080) (N=52) | 160 mg Elinzanetant (BAY3427080) (N=52)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (4) | 2 (2) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 4 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Viral sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 1 (2) | 3 (3) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
Headache (Nervous system disorders) | 6 (8) | 3 (3) | 2 (2) | 6 (7) | 4 (6)
Somnolence (Nervous system disorders) | 1 (2) | 3 (3) | 1 (1) | 2 (2) | 6 (6)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is required to postpone communication of results until a joint, multicenter publication of the multicenter study has occurred, or the sponsor confirms that no joint publication will be prepared, or 18 months since completion of the data analysis have passed. The sponsor can review planned publications for up to 60 days and request reasonable amendments. The review period can be extended by up to 6 months in case a patent application is planned.

DOCUMENTS (2):
  • Study Protocol (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT03596762/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03596762/SAP_001.pdf